# Reporting and Analysis Plan

**Study ID:** 117172

**Official Title of Study:** Reporting and Analysis Plan for ING117172 A Phase IIIb, randomized, open-label study of the safety and efficacy of dolutegravir/abacavir/lamivudine once daily compared to atazanavir and ritonavir plus tenofovir/emtricitabine once daily in HIV-1 infected antiretroviral therapy naïve women

**US IND:** 114,820

**EudraCT:** 2012-005823-34

**Date of Document:** 19-Aug-2022

# The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| randomized, open-label study<br>dolutegravir/abacavir/lamivud<br>atazanavir and ritonavir plus to | | Reporting and Analysis Plan for ING117172 A Phase IIIb, randomized, open-label study of the safety and efficacy of dolutegravir/abacavir/lamivudine once daily compared to atazanavir and ritonavir plus tenofovir/emtricitabine once daily in HIV-1 infected antiretroviral therapy naïve women |
|---|---|---|
| <b>Compound Number</b> | : | GSK1349572+GR109714+GI265235 (GSK2619619) |
| Effective Date | : | Refer to the document date |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Reports for Protocol ING117172.
- This RAP is intended to describe all the planned analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.
- The purpose of RAP Amendment 01 (to the originally approved RAP dated 20-OCT-2015) is to provide details on the Final (End of Study) analysis.

### **Author's Name and Functional Area:**

| Author | Date |
|---------------------------------------|-------------|
| Lead | |
| PPD | 01.4. 2022 |
| Associate Statistician, Biostatistics | 01-Aug-2022 |

# **RAP Team Reviews:**

# **RAP Team Review Confirmations (Vault TMF):**

| Reviewer | Date |
|---------------------------------------------------|-------------|
| PPD | 19-Aug-2022 |
| Principal Programmer/ Analyst, Biostatistics, GSK | |
| PPD | 19-Aug-2022 |
| Clinical Science Lead, ViiV | |
| PPD | 19-Aug-2022 |
| Safety Lead, GSK | |
| PPD | 19-Aug-2022 |
| Clinical Development Leader, ViiV | |
| PPD | 19-Aug-2022 |
| Clinical Development Manager, ViiV | |
| PPD | 19-Aug-2022 |
| Study Delivery Lead, GSK | |

# **Approval (Vault TMF):**

| Approver | |
|-----------------|------|
| PPD | |
| Manager, Statis | tics |

Copyright 2022 ViiV Healthcare and the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# CONFIDENTIAL

# The GlaxoSmithKline group of companies

ING117172

The main changes included in RAP Amendment 01 are:

Addition of Appendix 13 (Section 12.13) to provide additional details of the planned analyses and data displays for ING117172 Final/End of Study (EoS) reporting.

Appendix 14 (List of data displays) updated to reflect the updates to the EoS analyses in Appendix 13.

# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | CHRONOLOGY | 6 |
| 2. | REPORTING & ANALYSIS PLAN SYNPOSIS | 6 |
| 3. | SUMMARY OF KEY PROTOCOL INFORMATION | Q |
| J. | 3.1. Changes to the Protocol Defined Statistical Analysis Plan | |
| | 3.2. Study Objective(s) and Endpoint(s) | |
| | 3.3. Study Design | |
| | 3.4. Statistical Hypotheses | 10 |
| 4. | PLANNED ANALYSES | 10 |
| →. | 4.1. Interim Analyses | |
| | 4.2. Final Analyses | |
| | • | |
| 5. | ANALYSIS POPULATIONS | |
| | 5.1. Protocol Deviations | 12 |
| 6. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 40 |
| | CONVENTIONS | 12 |
| 7. | STUDY POPULATION ANALYSES | 14 |
| | 7.1. Overview of Planned Analyses | |
| | • | |
| 8. | PRIMARY STATISTICAL ANALYSES | 15 |
| | 8.1. Efficacy Analyses | 15 |
| | 8.1.1. Overview of Planned Efficacy Analyses | 16 |
| | 8.1.2. Planned Efficacy Statistical Analyses | 17 |
| 9. | SECONDARY STATISTICAL ANALYSES | _ |
| | 9.1. Efficacy Analyses | |
| | 9.1.1. Overview of Planned Efficacy Analyses | |
| | 9.2. Safety Analyses | |
| | 9.2.1. Overview of Planned Analyses | |
| | 9.2.2. Planned Safety Statistical Analyses | 24 |
| 10. | OTHER STATISTICAL ANALYSES | 26 |
| | 10.1. Health Outcomes | 26 |
| | 10.2. Virology | 27 |
| 11. | REFERENCES | 28 |
| 12 | APPENDICES | 29 |
| | 12.1. Appendix 1: Protocol Deviation Management and Definitions for | Per |
| | Protocol Population | |
| | 12.1.1. Exclusions from Per Protocol Population | |
| | 12.2. Appendix 2: Time & Events | 31 |
| | 12.2.1. Protocol Defined Time & Events | |
| | 12.3. Appendix 3: Assessment Windows | |
| | 12.3.1. Definitions of Assessment Windows for Analyses | 34 |

# CONFIDENTIAL

ING117172

| 12.4. | Appendix 4: Treatment States & Phases | 34 |
|--------|--------------------------------------------------------------|----|
| | 12.4.1. Treatment Phases | 34 |
| | 12.4.2. Treatment States | 34 |
| | 12.4.3. Treatment Phases and States | 37 |
| 12.5. | Appendix 5: Data Display Standards & Handling Conventions | 38 |
| | 12.5.1. Study Treatment & Sub-group Display Descriptors | 38 |
| | 12.5.2. Baseline Definition & Derivations | |
| | 12.5.3. Reporting Process & Standards | 38 |
| 12.6. | Appendix 6: Derived and Transformed Data | |
| | 12.6.1. General | 40 |
| | 12.6.2. Study Population | |
| | 12.6.3. Safety | 43 |
| | 12.6.4. Efficacy | |
| | 12.6.5. Viral Genotyping and Phenotyping | |
| | 12.6.6. Health outcomes | |
| 12.7. | Appendix 7: Premature Withdrawals & Handling of Missing Data | |
| | 12.7.1. Premature Withdrawals | |
| | 12.7.2. Handling of Missing Data | |
| 12.8. | Appendix 8: Values of Potential Clinical Importance | |
| 12.9. | Appendix 9: Examination of Covariates and Subgroups | |
| | 12.9.1. Handling of Covariates, Subgroups & Other Strata | |
| 12.10. | Appendix 10: Model Checking and Diagnostics for Statistical | |
| | Analyses | 55 |
| | 12.10.1. Statistical Analysis Assumptions | |
| 12.11. | Appendix 11: Snapshot | |
| | Appendix 12: Abbreviations & Trade Marks | |
| | 12.12.1. Abbreviations | |
| | 12.12.2. Trademarks | 61 |
| 12.13. | Appendix 13: Final (End of Study) Analysis | |
| | 12.13.1. Study Phases | |
| | 12.13.2. Analysis Populations for the Continuation Phase | |
| | 12.13.3. Study Population | |
| | 12.13.4. Safety Analysis | |
| | 12.13.5. Efficacy Analysis | |
| | 12.13.6. Virology Analysis | |
| | 12.13.7. COVID-19 Analysis | |
| | 12.13.8. List of Data Displays for Final (End of Study) | |
| 12.14. | Appendix 14: List of Data Displays | |
| | 12.14.1. Data Display Numbering | |
| | 12.14.2. Mock Example Shell Referencing | |
| | 12.14.3. Deliverable | |
| | 12.14.4. Study Population Tables | |
| | 12.14.5. Efficacy Tables | |
| | 12.14.6. Efficacy Figures | |
| | 12.14.7. Safety Figures | |
| | 12.14.8. Health Outcomes Tables | |
| | 12.14.9. Virology Tables | |
| | 12.14.10. Safety Tables | |
| | 12.14.11.ICH Listings | |
| | 12.14.12.Non-ICH Listings | |
| 12.15. | Appendix 15: Example Mock Shells for Data Displays | |

# 1. CHRONOLOGY

| Main RAP | 21-OCT-2015 | SF_1 00 Reporting and Analysis Plan |
|---|---|---|
| | | (RAP)_ARIA_21Oct2015_v1 (Week 48 Interim Analysis) |
| Amendment 1 | DD-MMM-YYYY | Appendix 13 added to provide details of the Analysis Plan |
| | | for the Final (End of Study) Analysis. |

# 2. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP describes all the planned analyses and outputs required for the Clinical Study Report(s) for Protocol ING117172. |
| Protocol | This RAP is based on protocol amendment 03 [Dated: 19/JUN/2018 of study ING117172 (GSK Document No.:2013N161649_01) and eCRF Version 9.0. |
| Primary<br>Objective | To demonstrate the non-inferior antiviral activity of DTG/ABC/3TC FDC once daily compared to ATV+RTV+TDF/FTC FDC each administered once daily over 48 weeks in HIV-1 infected ART naïve women. |
| Primary<br>Endpoint | The proportion of subjects with plasma HIV-1 RNA <50 copies/mL at Week 48 using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure) for the ITT-E population. |
| Study<br>Design | A 48 week Phase IIIb randomized, open-label, active-controlled, multicenter, parallel group, non-inferiority study. |
| | The study will be conducted in approximately 474 HIV-1 infected ART-naïve women. |
| | Subjects will be randomized 1:1 to receive a FDC of DTG 50mg/ ABC 600mg/<br>3TC 300mg once daily or ATV 300mg plus RTV 100mg and TDF 300mg/ FTC 200mg FDC each administered once daily. |
| | <ul> <li>Randomization will be stratified by Screening plasma HIV-1 RNA (≤100,000 copies/mL [c/mL] or &gt;100,000 c/mL) and CD4+ cell count (≤350 cells/mm3 or &gt;350 cells/mm3).</li> </ul> |
| | The study will comprise a Screening Phase (approximately 14-28 days), a Randomized Phase (48 weeks), and a Continuation Phase. |
| | No dose reductions, modifications in dosage, or changes in the frequency of dosing of any components of each regimen will be allowed in this study. |
| Planned<br>Analyses | The main analysis will be conducted to evaluate the primary objective of the protocol when all subjects have completed their Week 48 visit. A final analysis will be conducted when all subjects have completed the study. Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications and pricing reimbursement dossiers. |
| Analysis<br>Populations | The Intent-to-Treat Exposed (ITT-E) Population will be used for summaries of efficacy and study population. The Safety Population will be used for |

| Overview | Key Elements of the RAP |
|---|---|
| | summaries of safety. |
| | A 'Per-Protocol' Population and an Intent-to-Treat Population will be used to evaluate efficacy in sensitivity analyses. |
| | Separate populations for virology analyses will also be defined. |
| Hypothesis | This study is designed to show that the antiviral effect of the DTG/ABC/3TC FDC administered once daily is non-inferior to once daily ATV+RTV+TDF/FTC FDC. Non-inferiority can be concluded if the lower bound of a two-sided 95% confidence interval for the difference in response rates between the two treatment arms is greater than -12%. |
| Primary<br>Analyses | The primary endpoint will be analyzed using a Cochran-Mantel-Haenszel stratified analysis, adjusting from baseline stratification factors. A point estimate and corresponding 95% confidence interval will be constructed for the adjusted difference in response rates between DTG and ATV treatment groups. |
| | The primary analysis will be based on the ITT-E population using the Snapshot dataset. The primary comparison will be made at a one-sided 2.5% level of significance. |
| Secondary | Proportion of subjects with plasma HIV-1 RNA <50 and <400 c/mL over time |
| Analyses | Absolute values and changes from baseline in plasma HIV-1 RNA over time |
| | Absolute values and changes from baseline in CD4+ cell counts over time |
| | Incidence of HIV-1 disease progression |
| | Safety data will be presented in tabular format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |
| | Change from baseline in fasting lipids. |

# 3. SUMMARY OF KEY PROTOCOL INFORMATION

# 3.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in protocol amendment 1 (Dated: 12/AUG/2013).

# 3.2. Study Objective(s) and Endpoint(s)

| Objectives | | Endpoints | |
|---|---|---|---|
| Pri | Primary Objectives | | mary Endpoints |
| • | To demonstrate the non-inferior antiviral activity of DTG/ABC/3TC FDC once daily compared to ATV+RTV+TDF/FTC FDC each administered once daily over 48 weeks in HIV-1 infected ART naïve women. | • | The primary endpoint for this study will be the proportion of subjects with plasma HIV-1 RNA <50 copies/mL at Week 48 using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure) for the ITT-E population |
| Se | condary Objectives | Se | condary Endpoints |
| • | To evaluate the antiviral and immunological activity and incidence of disease progression (HIV-associated conditions, AIDS and death) of DTG/ABC/3TC FDC once daily compared to ATV+RTV+TDF/FTC FDC once daily over time; To compare the safety, tolerability, and laboratory parameters of DTG/ABC/3TC FDC once daily to ATV+RTV+TDF/FTC FDC once daily | • | Proportion of subjects with plasma HIV-1 RNA <50 and <400 c/mL over time; Absolute values and change from Baseline in plasma HIV-1 RNA over time; Absolute values and changes from Baseline in CD4+ cell counts over time; Incidence of disease progression (HIV-associated conditions, AIDS and death). Incidence and severity of AEs and laboratory abnormalities; Absolute values and changes over time in laboratory parameters; |
| | over time; | • | Proportion of subjects who discontinue treatment due to AEs; Change from Baseline in fasting lipids and glucose; |
| • | To assess the development of viral resistance in subjects who meet confirmed virologic withdrawal criteria; | • | Incidence of treatment-emergent genotypic and phenotypic resistance in subjects who meet confirmed virologic withdrawal criteria. |
| • | To evaluate renal markers (in urine and blood), and bone markers (in blood) in subjects treated with DTG/ABC/3TC FDC compared to ATV+RTV+TDF/FTC FDC; | • | Changes from Baseline in renal and bone markers. |
| • | To assess treatment satisfaction, and change in health-related quality-of-life for subjects treated with DTG/ABC/3TC FDC compared to ATV+RTV+TDF/FTC FDC; | • | Change from Baseline in health related quality of life using SF-12 at Week 48. Treatment satisfaction for subjects treated with DTG/ABC/3TC FDC once daily and those treated with ATV+RTV+TDF/FTC FDC once daily at weeks 4, 12, 24, and 48 (or withdrawal from the study). |

| Objectives | Endpoints |
|---|---|
| To evaluate the effect of patient characteristics (i.e., demographic factors, HIV-1 subtype, Baseline CD4) on response to DTG/ABC/3TC FDC compared to ATV+RTV+TDF/FTC FDC over time. | Proportion of subjects with plasma HIV-1 RNA <50 c/mL over time by subgroups. |

# 3.3. Study Design



# 3.4. Statistical Hypotheses

This study is designed to show that the antiviral effect of the DTG/ABC/3TC FDC administered once daily is non-inferior to once daily ATV+RTV+TDF/FTC FDC.

Non-inferiority can be concluded if the lower bound of a two-sided 95% confidence interval for the difference in response rates between the two treatment arms is greater than -12%. If r<sub>d</sub> is the response rate on DTG/ABC/3TC FDC and r<sub>a</sub> is the response rate on ATV+RTV+TDF/FTC FDC then the hypotheses can be written as follows:

H0: 
$$r_d - r_a \le -12\%$$
 H1:  $r_d - r_a \ge -12\%$ .

### 4. PLANNED ANALYSES

# 4.1. Interim Analyses

The main analysis will be conducted to evaluate the primary objective of the protocol when all subjects have completed their Week 48 visit. Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications.

The planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the Week 48 visit as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

# 4.2. Final Analyses

A final End-of-Study analysis will be conducted when all subjects have completed the study.

Details of which outputs will be produced at Week 48 and End of Study can be found in Section 12.14.

# 5. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Screened | <ul> <li>Comprised of all subjects screened for inclusion in the study.</li> <li>Subjects may be re-screened once, for which they will receive a new subject number.</li> <li>Only the latest re-screening data will be included in the screening population summaries/analyses but all screening data will be listed.</li> </ul> | Study Population |
| Safety | Comprise of all subjects who receive at least one dose of study treatment. | Safety |
| | This population will be based on the treatment<br>the subject actually received. If a subject<br>receives treatment differing from that assigned<br>by the randomization schedule (for either a<br>portion of or the entire time on study), they will<br>be analysed based on the treatment taken for<br>the majority of study participation. | |
| Intent-To-Treat (Exposed) | Comprise of all randomized subjects who receive at least one dose of study treatment. | Efficacy Chudu Papulation |
| | This population will be based on the treatment to which the subject was randomized. | <ul><li>Study Population</li><li>Health Outcomes</li></ul> |
| | Any subject who receives a treatment randomization number will be considered to have been randomized. | |
| Intent-To-Treat | Comprise of all randomized subjects. | Efficacy (sensitivity analyses) |
| | This population will be based on the treatment to which the subject was randomized. | analyses) |
| | Any subject who receives a treatment randomization number will be considered to have been randomized. | |
| Per-Protocol | Comprise of all subjects in the ITT-E population with the exception of major protocol violators, e.g. violations which could affect the assessment of antiviral activity. | Efficacy (sensitivity analyses) |
| | Protocol deviations that would exclude subjects from the PP population are defined in Section 5.1(Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population). | |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Viral Genotypic | Comprise of all subjects in the ITT-E population with available On-treatment genotypic resistance data at the time confirmed virologic withdrawal criterion is met (see protocol, Section 4.5.1). | Genotypic |
| Viral Phenotypic | Comprise of all subjects in the ITT-E population with available On-treatment phenotypic resistance data at the time confirmed virologic withdrawal criterion is met (see protocol, Section 4.5.1). | Phenotypic |

#### 1. NOTES:

 Please refer to Appendix 14: List of Data Displays which details the population to be used for each displays being generated.

### 5.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population)].
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - O Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 6. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are no planned adjustments made for multiple centres in this study.
- There are no planned adjustments for multiple comparisons or multiplicity.
- There are no PK analyses planned in this study.

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

# Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 12.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 12.2 | Appendix 2: Time & Events |
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Treatment States and Phases |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |
| 12.9 | Appendix 9: Examination of Covariates and Subgroups |
| 12.10 | Appendix 10: Model Checking and Diagnostics for Statistical Analyses |
| 12.11 | Appendix 11: Snapshot |
| 12.12 | Appendix 12: Abbreviations & Trade Marks |
| 12.13 | Appendix 13: Final (End of Study) Analysis |
| 12.14 | Appendix 14: List of Data Displays |
| 12.15 | Appendix 15: Example Mock Shells for Data Displays |

# 7. STUDY POPULATION ANALYSES

# 7.1. Overview of Planned Analyses

The study population analyses will be based on the ITT-E population, and will include a total column, unless otherwise specified. All displays are for the randomised phase only, unless otherwise stated.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Display | y's Generated |
|---|---|---|
| | Table | Listing |
| Randomisation | | • |
| Randomisation | | Υ [1] |
| Subject Disposition | | • |
| Study Populations [2] | Y | Y [3] |
| Study Recruitment [2] | | Y |
| Age Categories | Y | |
| History of Rescreened Subjects | | Υ |
| Reasons for Screen Failure [2] | Y | Υ |
| Subject Disposition | <b>Y</b> [4,9] | |
| Reasons for Withdrawal by Visit | Υ | Y |
| Study Visit Dates | | Y |
| Important Protocol Deviations | Y | Y |
| Deviations leading to exclusion from PP | Y | Y |
| Inclusion and Exclusion Criteria Deviations | | Y |
| Demography | | • |
| Demographic Characteristics <sup>[10]</sup> | Y | Y |
| Race & Racial Combinations <sup>[11]</sup> | Y | Y |
| Hepatitis Status | Y | Y |
| CDC Classification of HIV infection | Y | Υ |
| HIV Risk Factor | Y | Υ |
| Cardiovascular Risk Assessments at Day 1 | Y | Υ |
| Distribution of Quantitative Plasma HIV-1 RNA | Y | |
| Distribution of CD4+ Cell Counts | Y | |
| History of Cardiac Therapeutic Procedures | | Y |

| Display Type | Data Display | 's Generated |
|---|---|---|
| | Table | Listing |
| Medical Conditions, Concomitant Medications & Ar | tiretroviral Therapy | |
| Medical Conditions (Current and Past) [12] | Υ | <b>Y</b> [8] |
| Medical Conditions: Sub-conditions (Current/Past) [12] | Υ | <b>Y</b> [8] |
| Concomitant Medications (non-ART) | Υ[5] | Υ[6,8] |
| Prior and Concomitant ART Medications | | <b>Y</b> [7,8] |
| Lipid Modifying agents (Baseline and Post-Baseline) | Y | |
| Other | | |
| IP Accountability [13] | | Y |

#### 1. NOTES:

- Y = Display Generated, T = Tables, L = Listings, IP = Investigational Product
- 1. One listing of subjects randomised but not treated, and one listing of planned and actual treatment strata.
- 2. All Subjects screened population.
- 3. Listing only includes those who were excluded from at least one population.
- 4. Randomised Phase only at Week 48 analysis; Combined Randomised Phase and Continuation Phase for End of Study analysis.
- 5. Three separate tables, summarised by Ingredient ATC Level 1, Ingredient combinations and Combination term ATC Level 1 (EG Includes single-ingredient medications with multi-ingredient medications labelled according to the sum of their ingredients, e.g., "TYLENOL Cold and Flu" would appear as "CHLORPHENAMINE MALEATE + DEXTROMETHORPHAN HYDROBROMIDE + PARACETAMOL + PSEUDOEPHEDRINE HYDROCHLORIDE" under the ATC headings for "Nervous System" and "Respiratory System" (the combination's ATC classifications).)
- One listing for concomitant non-ART medications and one listing showing the relationship between verbatim text, ingredient and ATC Level 1.
- 7. One listing for Prior ART, one listing for concomitant ART and one listing showing the relationship between verbatim text, ingredient, combination and ATC Level 4.
- 8. Repeated for subjects at Mexico sites who experienced an adverse event, at End of Study reporting only.
- 9. Subjects who have not been recorded as either completing or withdrawing from the study will be categorized as "Ongoing at time of the analysis" for summary purposes.
- 10. Age, ethnicity, weight and height collected at screening (Day 1 for height)
- 11. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 12. Medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
- 13. Dispensation information (dates and number of tablets dispensed and returned)

# 8. PRIMARY STATISTICAL ANALYSES

# 8.1. Efficacy Analyses

The primary efficacy analyses will be based on the Intent-To-Treat (Exposed) population, unless otherwise specified. Summaries will be presented by treatment group with no total column.

All displays are for the randomised phase only, unless otherwise stated.

# 8.1.1. Overview of Planned Efficacy Analyses

Table 3 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 3 Overview of Planned Efficacy Analyses

| Endpoints | St | ats Analy | sis | Sum | mary | Indiv | idual |
|---|---|---|---|---|---|---|---|
| | T | F | L | Т | F | F | L |
| Proportion of Subjects with Plasma HIV-1 RNA <50c/ml at Week 48 – Snapshot | | | | | | | |
| Primary Analysis | <b>Y</b> [1] | | | <b>Y</b> [2] | <b>Y</b> [3] | | <b>Y</b> [2] |
| Treatment Heterogeneity across randomization strata | Y | | | | | | |
| <50 c/mL by<br>Subgroups [4] | | | | Y | Y[5] | | |
| Proportion of subjects analysis | without v | virologic | (ERDF) o | or virologic/to | lerability (TRI | OF) failure – S | ensitivity |
| Kaplan-Meier estimates | | | | Y | | | |

#### 1. NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Generated using the 'Intent-to-Treat Exposed' (primary), 'Per-Protocol' and 'Intent-to-Treat' (sensitivity)
  populations.
- 2. Study outcomes (i.e., response below 50 c/mL, virologic failure or reason for no data in the window) based on the snapshot algorithm.
- 3. Line plots, with 95% confidence intervals, for the proportion of subjects below 50 c/mL by treatment group at each visit
- 4. Baseline demography (age, race, country, CDC), HIV-1 subtype, Baseline CD4 and Baseline viral load
- 5. Plot of 95% confidence intervals for the proportion of subjects below 50 c/mL by subgroup.

# 8.1.2. Planned Efficacy Statistical Analyses

# **Primary Statistical Analyses**

# **Endpoint**

 Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure) for the ITT-E population

### **Snapshot Dataset**

- The Snapshot algorithm treats all subjects without HIV-1 RNA data at the visit of interest (due
  to missing data or discontinuation of IP prior to the visit window) as non-responders, as well as
  subjects who switch their concomitant ART prior to the visit of interest in certain scenarios.
   Since changes in ART are not permitted in this protocol, all such subjects who change ART will
  be considered non-responders.
- Otherwise, virologic success or failure will be determined by the last available HIV-1 RNA assessment while the subject is On-treatment within the visit of interest analysis window (see Section 12.3.1)
- Full details of the Snapshot algorithm are in Appendix 11.

# **Model Specification**

- The primary endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for Baseline plasma HIV-1 RNA ( ≤ vs. >100,000 c/mL) and CD4+ cell count (≤350 cells/mm3 or >350 cells/mm3).
- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each of the following four Baseline analysis strata:
  - $\circ$  Plasma HIV-1 RNA  $\leq$  100,000 c/mL AND CD4+  $\leq$  350 cells/mm3
  - Plasma HIV-1 RNA ≤ 100,000 c/mL AND CD4+ > 350 cells/mm3
  - Plasma HIV-1 RNA > 100,000 c/mL AND CD4+ ≤ 350 cells/mm3
  - Plasma HIV-1 RNA > 100,000 c/mL AND CD4+ > 350 cells/mm3
- If n<sub>k</sub> is the number of DTG treated subjects, m<sub>k</sub> is the number of ATV treated subjects, and N<sub>k</sub> = n<sub>k</sub> + m<sub>k</sub> is the total number of subjects in the kth stratum, then the CMH estimate is given by

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where,

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and dk are estimates of the differences in response proportions between the

# **Primary Statistical Analyses**

two treatment arms, r<sub>d</sub>-r<sub>a</sub>, for the kth strata.

• The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\hat{\text{var}}(\hat{d}_{cmh})}$$

using the variance estimator, var(d<sub>cmh</sub>), given by [Sato, 1989], which is consistent in both sparse data and large strata. The full equation for this variance estimate is provided in Section 12.6.4.

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of responders between each treatment group (DTG – ATV) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval
  (CI) for the CMH adjusted difference in the proportion of patients who respond in the DTG
  group minus the proportion of patients who respond in the ATV group is greater than -12%.

# Sensitivity and Supportive Statistical Analyses

- 1. Treatment Heterogeneity across randomization strata:
  - The weighted least squares chi-squared statistic [Fleiss, 1981] will be used to test for oneway homogeneity across the levels of each categorical variable, with each categorical variable considered separately.
  - Following Lui and Kelly [Lui, 2000] ½ will be added to each cell in any strata for which the stratum-specific rate estimates of either rd or ra are zero or one, and tests will be onesided.
  - Any heterogeneity found to be statistically significant will be explored and if necessary
    results will be reported for each level of the categorical variable. Investigation of
    heterogeneity will be confined to the primary. Tests of homogeneity will be assessed at the
    one-sided 10% level of significance.
- 2. Per-protocol population analysis:
  - To assess the impact of major protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis. If both analyses show non-inferiority then the hypothesis that the antiviral effect of treatment with DTG/ABC/3TC FDC is superior to treatment with ATV+RTV+TDF/FTC FDC will be tested at the two-sided 5% level of significance. Superiority will be declared if the lower end of the confidence interval is above 0% for the ITT-E population analysis. If superiority is declared the p-value for superiority will also be calculated.
- 3. Intent-to-Treat population analysis:
  - Statistical analysis will be repeated using the Intent-to-Treat population and compared for consistency with the results from the ITT-E and PP populations.
  - In this analysis, subjects randomised but not exposed to study treatment will be classified
    as non-responders, which therefore address any selection bias that may occur given the
    open-label study design.

### **Sensitivity and Supportive Statistical Analyses**

- 4. Exploration of Subgroups:
  - A simple analysis for all the subgroups listed in Section 12.9.1 will be performed. This will show the proportion of subjects with plasma HIV-1 RNA <50 c/mL at the time of analysis (Week 48) based on the SNAPSHOT algorithm and will be presented by treatment group.
  - Unadjusted difference in proportions between treatment groups and corresponding twosided 95% CI will also be presented by treatment and subgroup, and a 95% CI for the (unadjusted) treatment difference in each subgroup. These results will also be presented graphically.
  - If the basic summary suggests an interaction, then a corresponding summary of study outcomes (i.e., response below 50 c/mL, virologic failure or reason for no data in the window) by subgroup will be produced.

Note: These subgroup analyses will be exploratory and likely underpowered so that interpretation may therefore focus on point estimates as well as the lower bounds of 95% CIs for the treatment differences and response rates. Additionally, multiple comparisons are being made which inflates the risk of false positive findings. Therefore, if consistent findings across the multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding of non-inferiority.

- 5. Proportion of subjects without virologic (ERDF) or virologic/tolerability (TRDF) failure:
  - Estimated using the Kaplan-Meier nonparametric method based on the time to Confirmed Virologic Withdrawal (CVW) or treatment related/efficacy related discontinuation (i.e., drugrelated AE, protocol defined safety stopping criteria, or lack of efficacy)
  - Subjects who have not met CVW criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment/lack of efficacy, will be censored.
  - The estimate of the standard error used to derive confidence intervals for the difference in proportions between treatment groups will be based on Greenwood's formula [Kalbfleisch, 1980]
  - The estimated proportion of subjects without Confirmed Virologic Withdrawal and not discontinued due to treatment related/efficacy related reasons at Week 48 will be presented by treatment group, along with estimated difference in proportions between treatment groups and its associated two-sided 95% CI.
  - The proportion of subjects with Confirmed Virologic Withdrawal will be summarized by visit.

# 9. SECONDARY STATISTICAL ANALYSES

# 9.1. Efficacy Analyses

# 9.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the Intent-To-Treat (Exposed) population, unless otherwise specified. All displays are for the randomised phase only, unless otherwise stated.

Table 4 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 4 Overview of Planned Efficacy Analyses

| Endpoints | | | Δ | bsolu | te | | | | Cł | ange | from | Basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | _ | F | Ш | Т | F | F | Ш | Т | F | Ш | Τ | F | F | L |
| Plasma HIV-1 RNA Ove | r Tim | е | | | | | | | | | | | | |
| Observed | | | | Υ | | <b>Y</b> [1] | Υ | | | | Υ | | | |
| <b>Proportion of Subjects</b> | with I | Plasm | a HIV | -1 RN | A <400 | 0 & <5 | 0 сорі | ies/ml | L - Sn | apsho | ot | | | |
| <50 c/mL by Visit | | | | <b>Y</b> [2] | | | | | | | | | | |
| <400 c/mL by Visit | | | | Υ | | | | | | | | | | |
| <400 c/mL Outcomes | | | | Υ | | | Υ | | | | | | | |
| Confirmed Virologic Wi | thdra | wal (C | CVW) | | | | | | | | | | | |
| CVW by Visit | | | | Υ | | | Υ | | | | | | | |
| HIV-1 RNA distribution<br>at time of suspected<br>and confirmed<br>Virologic withdrawal | | | | Y | | | | | | | | | | |
| CD4+ Cell Counts Ove | r Time | 9 | | | | | | | | | | | | |
| CD4+ Observed | | | | Υ | | | Υ | | | | Υ | | | Υ |
| Post-baseline HIV-1 Dis | ease | Prog | essio | n <sup>[3]</sup> | | | | | | | | | | |
| HIV Conditions including Recurrences | | | | Υ | | | Y | | | | | | | |
| HIV Conditions excluding Recurrences | | | | Y | | | | | | | | | | |
| HIV Disease<br>Progressions | | | | Υ | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

- 1. Individual plasma profiles
- 2. Repeated for End of Study using Observed data.
- 3. HIV disease progressions categories: CDC Category A at baseline to CDC Category B event; CDC Category A at baseline to CDC Category C event; CDC Category B at baseline to CDC Category C event; CDC Category C at baseline to new CDC Category C event and CDC Category A, B or C at baseline to death.

# 9.2. Safety Analyses

# 9.2.1. Overview of Planned Analyses

The safety analyses will be based on the Safety population, presented by treatment group with a total column unless otherwise specified.

The observed case (OC) dataset will be used, which contains the data that is available at a particular timepoint, with no imputation for missing values, unless otherwise stated.

All displays are for the randomised phase only, unless otherwise stated.

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Endpoint | | Ab | solut | е | Cha | nge fro | m Bas | eline | Max Post BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summ | mmary Individual | | Summary Individual | | | | Sum | mary | Individual | | |
| | Т | F | F | L | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | | | | | |
| Extent of Exposure | <b>Y</b> [1] | | | Y[2,14] | | | | | | | | |
| Adverse Events[3] | | | | | | | | | | | | |
| All AEs by SOC and Toxicity <sup>[5]</sup> | Y | | | <b>Y</b> [4] | | | | | | | | |
| Common AEs by freq | Υ | <b>Y</b> [<br>16] | | | | | | | | | | |
| Common Grade 2-4<br>AEs [6] | Υ | | | | | | | | | | | |
| All Drug-Related AEs by SOC and toxicity <sup>[5]</sup> | Y | | | | | | | | | | | |
| Common Drug-related<br>Grade 2-4 AEs <sup>[6]</sup> | Υ | | | | | | | | | | | |
| All SAEs by SOC | <b>Y</b> [1] | | | | | | | | | | | |
| Reason for<br>Considering as a<br>Serious Adverse Event<br>(FDA) | | | | Y | | | | | | | | |
| All Drug-Related SAEs | Υ | | | | | | | | | | | |

| Endpoint | | Ab | solut | е | Cha | nge fro | m Bas | eline | Max Post BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summ | ary | Ind | ividual | Sum | mary | Indiv | idual | Sum | mary | Indiv | idual |
| | Т | F | F | L | Т | F | F | L | Т | F | F | L |
| by SOC | | | | | | | | | | | | |
| Fatal SAEs | | | | Υ | | | | | | | | |
| Non-Fatal SAEs | | | | Υ | | | | | | | | |
| Withdrawal AEs | <b>Y</b> [1] | | | Υ | | | | | | | | |
| Common Non-Serious<br>AEs (FDAAA) | Y | | | | | | | | | | | |
| Number of<br>occurrences of<br>Common Non-serious<br>AEs by SOC<br>(EudraCT) | Υ | | | | | | | | | | | |
| Number of<br>occurrences of SAEs,<br>Drug-related AEs,<br>Fatal SAEs, and Drug-<br>related SAEs<br>(EudraCT) | Y | | | | | | | | | | | |
| AEs of Subjects at Mexico sites | | | | <b>Y</b> [18] | | | | | | | | |
| SAEs of Subjects at non-Mexico sites | | | | <b>Y</b> [18] | | | | | | | | |
| Pre-treatment AEs | | | | Υ | | | | | | | | |
| CV events | | | | Υ | | | | | | | | |
| PSRAE | | | | <b>Y</b> [17] | | | | | | | | |
| Laboratory Values Ove | r Time | | | | • | | • | | | | | |
| Clinical Chemistry | | | | Υ [7] | Υ | | | | | | | |
| Lipids (%) | | | | | Υ | | | | | | | |
| Fasted Lipid<br>(Triglycerides and<br>TC/HDL ratio) analysis | | | | | Υ[22] | | | | | | | |
| Hematology | | | | Υ [7] | Υ | | | | | | | |
| Urine Dipstick | | | | Υ [7] | Υ | | | | | Υ | | |
| Urine Concentration | | | | <b>Y</b> [7] | Υ | | | | | | | |
| Proteinuria shifts | | | | | | | | | | <b>Y</b> [9] | | |
| Liver Chemistries | | | | | | | | | | <b>Y</b> [8] | | |
| NCEP shifts in lipids | | | | | | | | | Υ | <b>Y</b> [10] | | |
| Total Cholesterol/HDL ratio | | | | | Υ | | | | | | | |
| Bone markers | | | | | Υ | | | | | | | |

| Endpoint | | Ab | solut | е | Char | nge fro | m Bas | eline | | Max P | ost BL | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summ | Summary Individual | | ividual | Summary Individual | | | | Sum | mary | Individual | |
| | T | F | F | L | Т | F | F | L | Т | F | F | L |
| Treatment Emergent La | aborator | у Тох | icitie | S <sup>[11]</sup> | | | | | | | | |
| Clinical Chemistry | | | | | | | | | Υ | | | |
| Hematology | | | | | | | | | Υ | | | |
| Other | | | | | | | | | | | | |
| ECG Findings | | | | <b>Y</b> [21] | | | | | | | | |
| Vital Signs | | | | Υ | | | | | | | | |
| Abacavir HSR | Υ | | | Υ [12] | | | | | | | | |
| Liver Assessment | | | | Υ [13] | | | | | | | | |
| Hepatobiliary<br>Abnormality criteria | <b>Y</b> [1,19] | | | | | | | | | | | |
| Columbia suicidality | Υ | | | Υ [15] | | | | | | | | |
| Subjects who became<br>Pregnant | | | | Y | | | | | | | | |
| Patient Profiles | | | | Y [20] | | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Randomisation Phase only at Week 48 analysis; Combined Randomisation Phase and Continuation Phase for End of Study analysis.
- 2. Includes reason for any dose change/interruption.
- 3. Adverse events will be coded using the MedDRA coding dictionary to give a preferred term and a system organ class. Summaries include only Post-baseline AEs with onset date up to cut-off date for reporting effort, listings include all AEs including those with onset pre- or post-treatment.
- 4. One listing of all AEs including verbatim text and preferred term, one showing the relationship between verbatim text, preferred term and SOC and another giving subject numbers for individual all treatment emergent AEs.
- 5. For AEs reported more than once by a subject, the most severe intensity will be included.
- 6. Common AEs are those with >5% incidence in either treatment group summarised by frequency.
- 7. Listings for subjects with abnormalities for potential clinical concern, defined as any Grade1-4 toxicity.
- 8. Scatter plot of baseline vs. maximum post-baseline for ALT. Scatter plot of maximum ALT vs. maximum Bilirubin.
- 9. Shift table summarising baseline vs. maximum post-baseline result for urine dipstick protein
- 10. Bar chart for LDL, HDL, TC, Trig and HDL/TC ratio.
- 11. Treatment Emergent Laboratory Toxicities See protocol Section 11.2, Appendix 2.
- 12. Separate listings for exposure to abacavir, history of drug allergies, family conditions, skin rash, symptoms, vital signs, individual symptoms and diagnostic category assignment.
- 13. Separate listings for time of event from trt, RUCAM score, biopsy, imaging, past/ current conditions & FU
- 14. Repeated for subjects at Mexico sites at End of Study reporting.
- 15. Includes Baseline and lists all visits for a subject who reports any ideation or behaviour at any visit.
- 16. Plots of incidence rates and relative risk with 95% CI for DTG vs. ATV.
- 17. Four PSRAE listings: Event and Description (Section 1- Section 2), Possible Cause (Section 3), Section 4 and Section 5- Section 8.
- 18. Only for End of Study reporting
- 19. One summary of subjects and another table showing Subject Ids.
- 20. Patient profiles for subjects meeting protocol defined liver stopping criteria and for patients with virologic failure. Patient profiles can also be provided for any other subjects, as necessary for medical review.

- 21. Only collected when a Cardivascular event occurs.
- 22. Primary analysis method is multiple imputation MAR. Repeated for sensitivity analyses using OC, LOCF and MMRM.

# 9.2.2. Planned Safety Statistical Analyses

### **Statistical Analyses**

### **Endpoints**

- Change from Baseline in fasted triglycerides at Week 48.
- Change from Baseline in fasted TC/HDL ratio at Week 48.

#### Covariates

- Baseline Plasma HIV-1 RNA (≤100,000 c/mL c/mL or >100,000 c/mL c/mL)
- Baseline CD4+ cell count (≤350 cells/mm3 cells/mm3 or >350 cells/mm3)
- Fasted triglycerides (mmol/L) and fasted TC/HDL measurements at Baseline, Week 12 and Week 36
- Age (>=50 or <50)

### **Data Handling**

- If a subject is on lipid-lowering therapy from Baseline, they will be excluded from the analysis.
- If a subject initiates lipid-lowering therapy during the study, all visits after that date will be set to missing.
- All other data remains as is (observed or missing).
- A multiple imputation technique will be used to deal with the missing data at week 48.

# **Model Specification**

- Multiple imputations will be drawn from a multivariate normal model for the data (including covariates) with a Markov Chain Monte Carlo (MCMC) approach used to estimate posterior distributions. A non informative prior will be used. A seed of 18 will be used in the SAS program. Where a subject has a monotone or non-monotone pattern of missingness, all of their missing observations can be imputed under this approach.
- Imputations will be drawn separately for subsets of subjects according to their treatment group, i.e., based on means and variance-covariances from the same treatment group (Missing At Random (MAR) approach) conditioning on observed covariates listed above. This will be known as the MAR method.
- The imputations will be carried out 1,000 times. An ANOVA will be performed on each datasets produced adjusting for baseline triglycerides (<5.65 mmol/L or ≥5.65 mmol/L) or TC/HDL ratio (<3.5 or ≥3.5), age, baseline plasma HIV-1 RNA and CD4+ cell count, regardless of their significance. PROC MIANALYZE in SAS will be used to combine the 1,000 estimated means and difference to produce one estimated mean with 95% CI and associated p-value for the adjusted mean difference between each treatment group at Week 48.</p>
- Interactions between treatment and each of the covariates will not be assessed.

# **Model Checking & Diagnostics**

Refer to Appendix 10: Model Checking and Diagnostics for Statistical Analyses.

### **Model Results Presentation**

 Adjusted means and corresponding standard error of means (SEs) will be presented for each treatment, together with estimated treatment difference (DTG – ATV) and corresponding 95% confidence interval and p-value.

# Statistical Analyses

# **Sensitivity Analyses**

- Two ANCOVA sensitivity analyses will be performed as follows:
  - using the standard Observed Case (OC) dataset, with no adjustment or imputation for withdrawing, initiating lipid-lowering agents or other missing data.
  - using the Lipid LOCF dataset (see Section 12.7.2.2), but also carrying forward the last observation to any missing visits.
- A MMRM analysis, with time crossed with treatment, age, baseline triglycerides (<5.65 mmol/L or ≥5 .65 mmol/L) or TC/HDL ratio (<3.5 or ≥3.5),baseline Plasma HIV-1 RNA and CD4+ cell count will also be conducted.

# 10. OTHER STATISTICAL ANALYSES

### 10.1. Health Outcomes

The Health Outcomes analyses will be based on the ITT(E) population and presented by treatment group unless otherwise specified.

All displays are for the randomised phase only, unless otherwise stated.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 6 Overview of Planned Health Outcome Analyses

| Endpoints | | | | Absolu | ıte | | | | | Char | nge from | Basel | ine | ne |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | Stats<br>Analysis | | Summary | | Individual | | | Stats<br>nalys | - | Summary | | Individual | |
| | Т | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| Quality of Life | | | | | | | | | | | | | | |
| SF-12 individual item scores by Visit - LOCF | | | | Y | | | | | | | | | | |
| SF-12 Total score, PCS<br>and MCS by Visit -<br>LOCF & Observed | | | | Y | | | | | | | <b>Y</b> [1] | | | |
| Treatment satisfaction | | | | | | | | | | | | | | |
| HIVTSQs individual item scores by Visit - LOCF | | | | Y | | | Υ | | | | | | | |
| HIVTSQs (at Weeks 4,<br>12, 24 and 48) - LOCF &<br>Observed | Υ[2] | | | | | | Υ | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Change from Baseline at Week 48
- 2. Separate summaries for Total score, Lifestyle/ease sub-score and General Satisfaction/Clinical sub-score.

#### Statistical Analyses

#### Endpoint(s)

- HIVTSQ total score
- HIVTSQ general satisfaction/clinical sub-score (items 1, 2, 3, 9, and 10)
- HIVTSQ lifestyle/ease sub-scores (items 4, 5, 6, 7 and 8)

#### Model Specification/Analysis Methodology

- Wilcoxon rank sum tests.
- No adjustment for multiplicity will be applied as these analyses will be considered exploratory.
- An LOCF dataset will be used as described in Section 12.7.2.2.
- The analysis will be repeated using an Observed Case dataset (as supportive analyses). No adjustment for

multiplicity will be applied as these analyses will be considered supportive.

#### **Model Results Presentation**

 Summary statistics will be presented by treatment group, with a p-value for the difference in the mean based on the Wilcoxon rank sum test.

# 10.2. Virology

The virology analyses of genotype data will be based on the Genotypic population, and analyses of phenotype data will be based on the Phenotypic population. Summaries will be presented by treatment group unless otherwise specified.

All displays are for the randomised phase only, unless otherwise stated.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 7 Overview of Planned Virology Analyses

| Endpoint | | Abso | olute | | | Change fro | m Baseline | ) |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | idual | Sum | mary | Individual | |
| | T | F | F | Ш | Τ | F | F | L |
| Genotypic resistance | | | | | | | | |
| Incidence of genotype at time of CVW <sup>[3]</sup> | <b>Y</b> [1] | | | Y | <b>Y</b> [1] | | | Y |
| Phenotypic resistance | | | | | | | | |
| Incidence of phenotype at time of CVW <sup>[3]</sup> | <b>Y</b> [2[ | | | Y | | | | |
| INI replication capacity at time of CVW[3] | | | | Y | | | | |
| Fold Change at time of CVW <sup>[3]</sup> | Y | | | | Y | | | |

- 1. NOTES:
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Separate outputs for INI and NRTI/NNRTI/PI mutations
- 2. Separate outputs by phenotypic cut-off and by number of drugs to which subjects are resistant.
- 3. Sample used for resistance testing is taken at the suspected visit date, and only tested once a subject confirms virological failure at a subsequent visit.

# 11. REFERENCES

- Anderson KM, Wilson PWF, Odell PM, Kannel WB. An updated coronary risk profile. A statement for health professionals. *Circulation*. 1991;83:356-362.
- Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.
- GlaxoSmithKline Document Number 2013N161649\_01. Study ID ING117172. A
  Phase IIIb, Randomized, open-label study of the safety and efficacy of
  dolutegravir/abacavir/lamivudine once daily compared to atazanavir and ritonavir
  plus tenofovir/emtricitabine once daily in HIV-1 infected antiretroviral therapy naïve
  women. Report Date 12-AUG-2013.
- Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). *JAMA*. 2001;285 (19):2486-2497.
- HIVTSQ user guidelines
- Kalbfleisch J.D., Prentice R.L. *The Statistical Analysis of Failure Time Data.* 1st ed. New York: John Wiley & Sons; 1980.
- Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, *Biometrics*, 2000;56:309-315.
- Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989;42:311-323.
- Ware, JE Jr. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. *Medical Care* 1996. 0025-7079. 34(3):220 Lippincott Williams & Wilkins, Inc.
- Wensing AM, Calvez V, Günthard HF et al. 2014 Update of Drug Resistance Mutations in HIV-1. *Topics in Antiviral Medicine* 2014; 22(3): 642-650.
- Woodcock A, Bradley C (2001). Validation of the HIV Treatment Satisfaction Questionnaire (HIVTSQ). Quality of Life Research. 10:517-531.
- Woodcock A, Bradley C (2006). Validation of the Revised 10-item HIV Treatment Satisfaction Questionnaire Status Version and New Change Version. Value in Health. 9:320-333.

# 12. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : Analysis Populations |
| Section 12.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 6 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 12.2 | Appendix 2: Time and Events |
| Section 12.3 | Appendix 3: Assessment Windows |
| Section 12.4 | Appendix 4: Treatment States & Phases |
| Section 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 12.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | • Virology |
| | Health outcomes |
| Section 12.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 12.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 12.9 | Appendix 9: Examination of Covariates and Subgroups |
| Section 12.10 | Appendix 10: Model Checking and Diagnostics for Statistical Analyses |
| Section 12.11 | Appendix 11: Snapshot |
| Other RAP App | |
| Section 12.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 12.13 | Appendix 13: Final (End of Study) Analysis |
| Section 12.14 | Appendix 14: List of Data Displays |
| Section 12.15 | Appendix 15: Example Mock Shells for Data Displays |

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 12.1.1. Exclusions from Per Protocol Population

Protocol deviations leading to exclusion from PP population are those deviations which

- may directly impact the efficacy endpoint of HIV-1 RNA; or
- lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the protocol deviations which, if they occur prior to an analysis timepoint of interest, will lead to exclusion of a subject from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. This review will occur before the clinical database has been frozen for analysis.

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 01 | Subject deviates from any inclusion or exclusion criteria, as recorded in the eCRF |
| 02 | Subject took/received incorrect IP, i.e., other than the one to which they were randomized for greater than 10% of the total time On-treatment |
| 03 | Interruption of IP for greater than 10% of the total time On-treatment, for reasons other than treatment-related adverse events/laboratory abnormalities, based on eCRF IP exposure forms (or CONMEDS eCRF forms for locally prescribed RTV during supply issues) |
| 04 | Prohibited medications: Receiving ART medication other than that prescribed/allowed by the study for a duration of >2 consecutive weeks or receiving non-ART medication that would potentially impact exposure or response to therapy with duration taken into consideration |
| 05 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF). |

# 12.2. Appendix 2: Time & Events

# 12.2.1. Protocol Defined Time & Events

| Procedures | Scree | D | | R | andom | ized Ph | ase | | Continuat | Withdra | Follo |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | na | ay<br>1 | | | | | | | ion | wal | w-up <sup>l</sup> |
| | | <b>'</b> | | <u> </u> | lala Via | :4- | | Canta | Phase <sup>k</sup> | | |
| | | | Wee | | inic Vis<br>Wee | | Wee | Conta ct at | Every 12<br>weeks | | |
| | | | vvee<br>k | Wee<br>k | vvee<br>k | Wee<br>k | vvee<br>k | Wk 8 | after | | |
| | | | 4 | 12 | 24 | 36 | 48 | 18, | Week 48 | | |
| | | | 7 | 12 | 24 | 30 | 70 | 30, | TICCK 40 | | |
| | | | | | | | | 42 <sup>r</sup> | | | |
| | | <u> </u> | CI | inical a | nd Oth | er Asse | ssmen | | | | |
| Written informed | Х | | | | | | | | | | |
| consent | | | | | | | | | | | |
| Inclusion/Exclusio | Х | X | | | | | | | | | |
| n criteria <sup>b</sup> | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | |
| Prior ART history | Х | | | | | | | | | | |
| Medical history <sup>c</sup> | | Х | | | | | | | | | |
| Current medical | | Х | | | | | | | | | |
| conditions | <u> </u> | | | | | | | | | | |
| HIV risk factors | | Х | | | | | | | | | |
| and mode of | | | | | | | | | | | |
| transmission | | | | | | | | | | | |
| CDC HIV-1 | Х | X | | | | | | | | | |
| classification | | | | | | | | | | | |
| HIV associated | | | X | X | Х | X | X | | Х | X | |
| conditions | | ļ., | | | | | | | | | |
| Cardiovascular | | X | | | | | | | | | |
| risk assessment <sup>d</sup> | | | | | | | | | | | |
| Columbia | | X | Х | Х | X | Х | Х | | Х | X | |
| Suicidality | | u | | | | | | | | | |
| Severity Rating Scale | | | | | | | | | | | |
| Concomitant | Х | Х | Х | Х | Χ | Х | Х | | Х | Х | Χ |
| medication | ^ | ^ | ^ | ^ | ^ | ^ | ^ | | ^ | ^ | ^ |
| Limited physical | Х | Х | Х | Х | Х | Х | Х | | Х | Х | χ |
| examination <sup>s</sup> | _ ^ | ^ | ^ | ^ | ^ | ^ | ^ | | ^ | ^ | _ ^ |
| 12-lead ECG <sup>t</sup> | Х | | | | | | | | | | |
| Adverse events | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Serious adverse | χj | X | X | X | X | X | X | X | X | X | X |
| events | ^, | ^ | ^ | ^ | _ ^ | ^ | ^ | ^ | ^ | Α | _ ^ |
| SF-12 <sup>w</sup> | | Х | | | Х | | Х | | | Х | |
| HIVTSQW | | | Χ | Χ | Х | | Χ | | | Х | |
| Confirm | | Χ | Х | Х | Х | Х | Χ | Х | Χ | | |
| understanding of | | | | | | | | | | | |
| study and | | | | | | | | | | | |
| management/toler | | | | | | | | | | | |
| ability of regimen | | | | | | | | | | | |
| | 1 | | П | Labor | ratory A | ssessn | nents | T | T | T | T |
| Plasma for HIV | Х | | | | | | | | | | |
| genotyping | <u> </u> | | | | | | | | | | |

| Procedures | Scree<br>n <sup>a</sup> | D<br>ay<br>1 | , | | | | | Continuat<br>ion<br>Phase <sup>k</sup> | Withdra<br>wal | Follo<br>w-up <sup>l</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | CI | inic Vis | its | | Conta | Every 12 | | |
| | | | Wee | Wee | Wee | Wee | Wee | ct at | weeks | | |
| | | | k | k | k | k | k | Wk 8 | after | | |
| | | | 4 | 12 | 24 | 36 | 48 | 18,<br>30,<br>42 <sup>r</sup> | Week 48 | | |
| Quantitative | Х | Х | Х | Х | Vn | Vn | vn | 72 | V/n | Х | |
| plasma HIV-1 RNA | | | | | Χn | Xn | Xn | | Χn | | |
| Lymphocyte subset | Х | X | Х | Х | Х | Х | Х | | Х | Х | Х |
| Plasma for storage <sup>e</sup> | Х | Х | Х | Х | Х | Х | Х | | Х | Х | Х |
| HLA-B* 5701 | Х | | | | | | | | | | |
| testing <sup>q</sup> | ^ | | | | | | | | | | |
| Clinical chemistry | Х | X | Х | X | X | X | X | | X | Χ | X |
| Hematology | Х | X | Χ | X | Χ | Χ | X | | Х | Χ | X |
| Fasting lipids and glucose <sup>f</sup> | | X | | Х | Х | Х | Х | | | | |
| Urinalysis and spot urine for protein analysis <sup>9</sup> | | Х | | | Х | | Х | | Хр | Χm | Х |
| Pregnancy test <sup>h</sup> | S | U | S | S | S | S | S | | S | S | |
| HBsAg and<br>hepatitis C<br>antibody | Х | | | | | | | | | | |
| Pharmacogenetic sample <sup>i</sup> | | Х | | | | | | | | | |
| Bone marker | | Х | | | Χ | | Χ | | | | |
| analytes (blood) <sup>v</sup> | | | | | | | | | | | |
| | | 1 | | | stigatio | | | 1 | | | |
| IVRS | Х | X | X | X | X | X | X | | Х | Х | Х |
| Dispense IP | | X | X | X | X | X | Χo | | Х | | |
| IP accountability (pill counts) | | | X | X | Х | X | X | | Х | X | |

- a. The 14-day Screening period maybe extended to 28 days. Randomization may occur as soon as all Screening results are available.
- Inclusion/exclusion criteria will be fully assessed at the Screening visit. Changes between the screening visit
  and the Day 1 visit should be assessed to ensure eligibility, including additional assessments performed at Day
  1.
- Full medical history will be collected. Targeted medical history assessments will include cardiovascular, metabolic (e.g., Type I or II DM), psychiatric (e.g, depression) and renal (e.g., nephrolithiasis, nephropathy, renal failure) disorders.
- d. Assessment for cardiovascular risk will include height, weight, blood pressure, smoking history, medical conditions, and family history of premature cardiovascular disease
- e. Plasma samples for storage will be collected at each visit for possible future analyses (including but not limited to HIV-1 RNA genotypic and phenotypic analyses, HIV-1 RNA levels, and immunological parameters). These samples will be used when needed such as when samples are lost or arrive at the laboratory unevaluable. Additionally, these samples will be used for genotypic and/or phenotypic analyses when subjects meet confirmed virologic withdrawal criteria.

- f. An overnight fast is preferred, however a minimum of a 6 hour fast is acceptable.
- g. A morning specimen is preferred.
- h. Pregnancy testing. Women of childbearing potential only. S=serum, U=urine. Remind females of reproductive potential of the need to avoid pregnancy while in study and adherence to the study's contraception requirements.
- Informed consent for optional pharmacogenetics (PGx) research must be obtained before collecting a sample.
   Collection of the PGx sample at Day 1 is preferred, however this sample may be collected at any time during the study.
- Only SAEs related to study participation or to a concomitantly administered GSK product will be collected between obtaining informed consent and administration of IP at Day 1.
- k. For subjects who completed randomized DTG/ABC/3TC FDC through Week 48 and entered into DTG/ABC/3TC FDC Continuation Phase: subjects completing the DTG/ABC/3TC FDC Continuation Phase must return to the clinic when transitioning to commercial supplies. Conduct study assessments as specified per the Week 36 schedule at this end of Continuation Phase visit.
- I. A Follow up visit may be conducted approximately 4 weeks after the last dose of study provided IP, and is required only if the subject has ongoing AEs or lab abnormalities at the last on study visit. The assessments performed should reflect what is considered medically necessary to assess the event(s).
- m. Conduct assessments at Week 48 OR at the Withdrawal visit for subjects who discontinue from the study prior to Week 48, but not both.
- n. Beginning at Week 24, subjects with plasma HIV-1 RNA ≥50 but <400 c/mL who elect to remain in study must return every 4-6 weeks for collection of samples for HIV-1 RNA determination and plasma for storage. Genotype and phenotype testing will only be performed with confirmed HIV-1 RNA ≥400 c/mL.
- o. For subjects receiving DTG/ABC/3TC FDC in Continuation Phase only
- p. Will be tested every 24 weeks (not every 12 weeks)
- q. Documentation that the subject had been screened for, and is negative for the HLA-B\*5701 allele is acceptable.
- r. Contacts at Week 8,18, 30 and 42 are mandatory but may be conducted as a telephone, clinic or home visit (or other type of visit as agreed with GSK).
- s. Limited physical examination to include blood pressure at Baseline (recorded in eCRF) for Framingham score assessment, and weight at each visit (recorded in eCRF at Baseline and on lab requisition at all visits) for determination of CrCL. Blood pressure to be measured after resting in a semi-supine position for at least 5 minutes.
- A 12-lead electrocardiograph (ECG) will be performed after resting in a semi-supine position for at least 5 minutes.
- u. On Day 1, the Columbia Suicidality Severity Rating Scale (conducted by voice response system) is to be administered prior to randomization.
- v. Blood sample for bone marker assessment. Only the result for 25 hydroxy-vitamin D will be reported to the investigator.
- w. SF-12 and HIV Treatment Satisfaction Questionnaire (HIVTSQ) is recommended to be administered at the beginning of the visit.

# 12.3. Appendix 3: Assessment Windows

Laboratory data, vital signs, ECGs, health outcomes assessments, and genotypic and phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database. The CVW algorithm will be derived using nominal CRF visit rather than using the assessment window defined below.

A window around a target Study Day will typically include all days from the midpoints between it and the target Study Days of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

### 12.3.1. Definitions of Assessment Windows for Analyses

| Analysis Set | Parameter | Target | Analysis | Analysis | |
|---|---|---|---|---|---|
| / Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | All | -28 | <=-4 | <=-4 | Screening |
| | | 1 | -3 | 1 | Day 1 |
| | | 29 | 2 | 56 | Week 4 |
| | | 85 | 57 | 126 | Week 12 |
| | | 169 | 127 | 210 | Week 24 |
| | | 253 | 211 | 294 | Week 36 |
| | | 337 | 295 | Date of Week<br>48 visit | Week 48 |
| | | 421 | Date of Week<br>48 visit +1 | 462 | Week 60 |
| | | 7*w + 1 | (7*w - 41) | (7*w + 42) | Week w<br>w = 72, 84,<br>96, |
| | | Study Day of last dose + 28 | > (Study Day of last dose + 1) | - | Follow-up |

#### 1. NOTES:

- For parameters which are not scheduled to be assessed at particular visits, the all- inclusive windows defined will still be used.
- Data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot).
   1.

# 12.4. Appendix 4: Treatment States & Phases

### 12.4.1. Treatment Phases

All displays are for the randomised phase only, unless specified otherwise.

Data collected from both arms up to and including the date of the Week 48 visit, or unscheduled Week 48 visit date, will be considered to be during the Randomised Phase of the Study.

Data collected from the DTG/ABC/3TC FDC arm after Week 48, or unscheduled Week 48 visit, to the end of the study will be considered to be during the Continuation Phase of the Study.

#### 12.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

# 12.4.2.1. Treatment States for Laboratory, HIV Associated Conditions, Vital Signs, ECGs, Health Outcomes and Genotypic and Phenotypic Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

#### 1. NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 12.4.2.2. Treatment States for AE Data

For adverse events, partial AE start date will use imputation as described in Section 12.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment unless an end date for the AE is provided which is before start of investigational product; in such a case the AE is assigned as Pre-treatment.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date <sup>&gt;</sup> AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

- If the study treatment stop date is missing, then any event with a start date on or after study treatment Start Date will be considered to be On-treatment.
- If the start date of the AE is after study treatment Stop Date but has been recorded as potentially related to study treatment, then it will be classified as On-treatment.
#### 12.4.2.3. Treatment States for Prior/Concomitant/Post-Therapy Medications Data

- Prior medications: Those taken (i.e., started) before the start date of investigational product.
- Concomitant medications: Those taken (i.e., started or continued) at any time between the start date and stop date of study treatment, inclusive. Prior medications that were continued during this period are also considered as concomitant medications.
- Post treatment medications: Those started after the stop date of study treatment. Concomitant medications that were continued during this period are also considered as post-treatment medications.

It will be assumed that medication has been taken on the date in which it is reported as started or stopped. For any medication starting on the same date as study treatment, it will be assumed that the medication was taken after the subject started taking study treatment.

ART medications will also be classified as prior, concomitant and/or post-treatment according with the following modifications:

- ART starting on study treatment stop date will be considered as only posttreatment and not concomitant. It is expected that after discontinuation of study treatment, a subject may immediately begin taking another ART.
- ART stopping on study treatment start date will only be considered as prior and not concomitant.
- Any ART entered on the Prior ART eCRF with partial end date will be assumed to have finished before Screeninig.

| | Pre-<br>treatment | | On-treatment | | Po | st-treatment | Prior | Conco-<br>mitant | Post |
|---|---|---|---|---|---|---|---|---|---|
| (a) | хх | | | | | | Υ | N | N |
| (b) | x | | ———х | | | | Υ | Υ | N |
| (c) | x | | | | | ———х | Υ | Υ | Υ |
| (d) | _ | | хх | | | | N | Υ | N |
| (e) | | بو | X | e | + | ———х | N | Υ | Υ |
| (f) | | IP Start Date | | IP Stop Date | IP Stop Date+1 | xx | N | N | Υ |
| (g) | ?x | art | | do | □ d | | Υ | N | N |
| (h) | ? | St | ———Х | St | Sto | | Y* | Υ | N |
| (i) | ? | <u> </u> | | Н | П | ———Х | Y* | Υ* | Υ |
| (j) | X | | | | | ? | Y | Y** | Y** |
| (k) | _ | | X | | | ? | N | Υ | Y** |
| (l) | | | | | | x? | N | N | Υ |
| (m) | ? | | | | | <del>?</del> | Y*** | Y*** | Y*** |
| (n) | x | Х | | | | | Υ | Υ | N |
| (o) | ? | Х | | | | | Y* | Υ | N |
| (p) | | Х | ———х | | | | N | Υ | N |
| (q) | | Х | | Х | | | N | Υ | N |
| (r) | | | | Х | | X | N | Υ | Υ |
| (s) | | | | Χ | | ? | N | Υ | Y** |
| (t) | | | | | Χ | ———х | N | N | Υ |
| (u) | | | | | Χ | ? | N | N | Υ |
| (v) | | | X | | Х | | N | Υ | Υ |

- 1. x = start/stop date of medication
- 2. ? = missing start/stop date of medication
- 3. \* If a medication is stopped On-treatment or Post-treatment and no start date is recorded it will be assumed that the medication was ongoing from the Pre-treatment phase
- 4. \*\* If a medication is started Pre-treatment or On-treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study
- 5. \*\*\* If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pretreatment phase to the Post-treatment phase

#### 12.4.3. Treatment Phases and States

On-treatment and Post-treatment assessments and events will be classified as occurring during the Randomized Phase or the Continuation Phase of the study as follow:

- If a subject did not enter the Continuation Phase, then any Post-treatment data will be assigned to the Randomized Phase.
- For subjects who did enter the Continuation Phase, any Post-treatment data will be assigned to the Continuation Phase.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

## 12.5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order [1] |
| Α | DTG/ABC/3TC FDC once daily | DTG/ABC/3TC | 1 |
| В | ATV +RTV +TDF/FTC FDC once daily | ATV +RTV +TDF/FTC | 2 |

#### NOTES:

# 12.5.2. Baseline Definition & Derivations

#### 12.5.2.1. Baseline Definitions

For all endpoints (unless stated otherwise) the baseline value will be the latest pre-dose assessment. This is generally expected to be from the Day 1 visit, although such values may be missing or unscheduled assessments may be performed before treatment start.

#### 12.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 12.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 12.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | Software |
| The currently supported versions of SAS software and TSCG will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : \ARPROD\GSK2619619\ING117172 |
| QC Spreadsheet : \ARPROD\ GSK2619619\ING117172\(Week48 or Final)\Documents | |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & | |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### **Reporting Process**

AdaM IG Version 1.0.

• For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for the Week 48 and end of study analyses.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Actual time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 12.3.1.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the T&E table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and
  in data listings, as well any algorithms that make use of additional data (e.g., SNAPSHOT).

#### **Reporting Standards**

### **Invalid Laboratory Assessments**

 Certain laboratory endpoints are required to be collected in a fasting state, i.e., glucose and lipids (triglycerides, total cholesterol, HDL, LDL). If these endpoints are collected in a nonfasting state, then the results will be excluded from summaries; such results will be included in data listings with the fasting status noted.

## **Descriptive Summary Statistics**

| Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
|------------------------------------------------------------|
| Categorical Data N, n, frequency, % |
| Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. |

# 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

### **Multiple Measurements at One Time Point**

- If after window assignment there are multiple valid (see Section 12.3) assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:
  - the assessment closest to the window target Study Day;
  - if there are multiple assessments equidistant from the target Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean
- Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, such valid assessments will be used when determining values of potential clinical concern for the 'any time On-treatment' time point, and for any algorithm that has specific rules for which observation to use (e.g., SNAPSHOT or LOCF).

#### **Study Day**

- Calculated as the number of days from initial study treatment start date :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date Treatment Start Date
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) + 1

Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Post-baseline

 Post-baseline refers to the combined time periods of On-treatment and Post-treatment. Postbaseline may be further specified according to phase of the study: Randomized or Continuation.

#### 12.6.2. Study Population

#### **Demographics**

#### Age

- Age, in whole years, will be calculated with respect to the subject's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied.
   Consequently, the age of the subject will not be calculated and will remain missing.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / Height (m)<sup>2</sup>

#### **Hepatitis Status**

- Hepatitis C status will be determined using antibody (IgM or IgG) and/or hepatitis C virus (HCV)
   RNA assessments performed during screening or during the conduct of the study.
- If both antibody and virus RNA assessments are available, then the latter will take precedence
  and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥43 IU/mL
  [≥1.63 log IU/mL]) or not.
- A subject will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen or detectable HBV DNA result during screening or during the conduct of the study.

# Framingham Risk Equation

• The predicted probability, p, for time (t = 4,...,12 years) of coronary heart disease according to the Framingham equation [Anderson, 1991] is:

$$p = 1 - \exp(-e^{u})$$
 where 
$$u = \frac{\log(t) - \mu}{\sigma}$$
 with 
$$\mu = 4.4181 + m$$
 and 
$$\sigma = \exp(-0.3155 - 0.2784 \times m)$$

The quantity m is calculated as

$$m = \begin{cases} a - 1.4792 \times \log(age) - 0.1759 \times I_d & \text{if male} \\ a - 5.8549 + 1.8515 \times \left[\log(age/74)\right]^2 - 0.3758 \times I_d & \text{if female} \end{cases}$$

where

#### **Demographics**

$$a = 11.1122 - 0.9119 \times \log(SBP) - 0.2767 \times I_s$$
$$-0.7181 \times \log(TC/HDL) - 0.5865 \times I_{IVH}$$

and

$$\begin{split} I_{d} &= \begin{cases} 1 & \text{if diabetic subject} \\ 0 & \text{otherwise} \end{cases} \\ I_{r} &= \begin{cases} 1 & \text{current or form er smoker} \\ 0 & \text{otherwise} \end{cases} \\ SBP &= \text{systolic blood pressure (mmHg)} \\ TC &= \text{total serum cholesterol} \\ HDL &= \text{serum HDL cholesterol} \\ I_{LVH} &= \begin{cases} 1 & \text{definite ECG for left ventricular hypertrophy} \\ 0 & \text{otherwise} \end{cases} \end{split}$$

with total cholesterol and HDL cholesterol measured in the same units.

- A subject is classified as diabetic if current or past is indicated in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or if baseline fasting glucose ≥7.00 mmol/L (126 mg/dL).
- Smoking status is collected in the eCRF on Day 1. A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used tobacco products within the previous 6 months.
- Definite ECG for left ventricular hypertrophy (LVH) is assessed based on current or past indication in the medical conditions eCRF for LVH.
- This calculation will not be performed for subjects who have indicated current or past
  myocardial infarction conditions on the eCRF. These subjects will not be included in summary
  statistics of risk, but will be counted in the highest category of risk in the summary by category.

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
  - In the situation where IP consists of more than one drug, the earliest start date and latest stop
- date will be used.
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- Missing Treatment Stop Date will be imputed, for purposes of calculating exposure, as the date of last visit or the recorded date of withdrawal/completion, whichever is earlier.
- An alternative calculation of exposure will be performed where the duration of any dosing interruptions based on eCRF data will be subtracted from the result above.
  - The ratio (percentage) of the actual exposure to the overall exposure (i.e. study

#### **Extent of Exposure**

treatment stop date – study treatment start date+1) will be used to define protocol deviation leading to exclusion from PP Population due to study treatment interruption (i.e. >10%).

 Due to local supply issues of RTV during the study, some subjects had to take locally prescribed RTV and this is reported on the CONEMDS eCRF rather than IP eCRF. When calculating interruptions, RTV records on the CONMEDS eCRF will be used in conjunction with the IP eCRF data.

## 12.6.3. Safety

#### **ECG Parameters**

#### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Adverse Events**

# **AE Severity – DAIDS Grading**

- The DAIDS grading for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria.

# **Laboratory Parameters**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

#### **Laboratory Parameters**

- $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
- Example 2: 1 Significant Digit = '> x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x 1

### Glomerular Filtration Rate (GFR)

• The Cockroft-Gault method will be used by the central laboratory to provide an estimate of GFR, in mL/min, as follows:

GFR = 
$$\frac{(140 - age) \times weight \times 88.4}{CRT_{\mu mol/L} \times 72} \times (0.85 \text{ if female})$$
$$= \frac{(140 - age) \times weight}{CRT_{mg/dL} \times 72} \times (0.85 \text{ if female})$$

where age (in years) and weight (in kg) are at time of assessment, and CRT $\mu$ mol/L is serum creatinine concentration in GSK standard units of  $\mu$ mol/L. CRTmg/dL is serum creatinine concentration in mg/dL, and CRT $\mu$ mol/L=88.4x CRTmg/dL.

#### Lab Toxicities - DAIDS Grading

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, as specified in the protocol.
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint | Above Midpoint |
|----------------|----------------|----------------|
| Fasted glucose | Hypoglycaemia | Hyperglycaemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

#### National Cholesterol Education Program (NCEP) Lipid Categories

• In addition to DAIDS toxicity scales (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001]

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |

| L | Laboratory Parameters | | | |
|---|---|---|---|---|
| | | 1.04 to <1.56 | 40 to <60 | Normal |
| | | ≥1.56 | ≥60 | High |
| | LDL Cholesterol | <2.59 | <100 | Optimal |
| | | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | | 4.14 to <4.92 | 160 to <190 | High |
| | | ≥4.92 | ≥190 | Very High |

#### Total Cholesterol / HDL Cholesterol Ratio

 When both total cholesterol and HDL cholesterol results are available from the same date for a subject, then the ratio will be calculated by dividing the total cholesterol result by the HDL cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------|--------------|
| Total Cholesterol | < 3.5 |
| / HDL Ratio | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥ 5 |

#### Other Safety Endpoints

### Columbia Suicide Severity Rating Scale (C-SSRS)

- Missing data will not have any imputation performed.
- Incomplete calls:
  - when no complete call is databased on the same day, the incomplete data will be used
  - when a complete call is databased on the same day, the data from the complete call will be used in the summaries.
- Duplicate calls:
  - If they occur on the same day, the latest entry will be used.
  - If they occur on different days, take the entry closest to the target visit date.

# **12.6.4.** Efficacy

#### **HIV-1 RNA**

#### **Snapshot (Missing, Switch or Discontinuation=Failure)**

- It is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- Virologic Success (e.g., <50 c/mL) or Virologic Failure within an analysis window (see Section 12.3.1) is typically determined by the last available HIV-1 RNA measurement in that window while the subject is On-treatment.
- When no HIV-1 RNA data is available within a window, a subject cannot be a Virologic

#### **HIV-1 RNA**

Success. Depending on the reason for lack of data, the subject will be classified as a Virologic Failure or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a subject withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a subject withdraw for reasons other than AE and was not suppressed at the time, they will be a Virologic Failure.

• For each scheduled assessment time, the snapshot response rate for a given threshold (e.g., <50 c/mL) is defined as:

Snapshot Rate = 
$$\frac{\text{Number of responders in that analysis window}}{\text{Number of subjects in the analysis population}}$$

 Full details of the algorithm, including the handling of special cases, are included in Section 12.11

#### Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For
  the purposes of summary statistics, such values will be replaced by the next value beyond the
  limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data
  listings will show the censored values as provided.

# Treatment (TRDF) and Efficacy Related (ERDF) Discontinuation = Failure

- The analysis of time to Confirmed Virologic Withdrawal or discontinuation due to treatment related reasons (i.e., drug-related AE, protocol defined safety stopping criteria, or lack of efficacy) will censor subjects who have not met CVW criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment. This will be the Treatment Related Discontinuation = Failure (TRDF) data.
- Subjects who have not met CVW criteria and are ongoing in the study, or who have discontinued for reasons other than lack of efficacy, will be censored in the analysis of the Efficacy Related Discontinuation = Failure (ERDF) data.

#### Variance Estimator of Cochran Mantel-Haenszel Risk Difference

• 
$$\operatorname{var}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{(\sum n_k m_k / N_k)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{(\sum W_k)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

## 12.6.5. Viral Genotyping and Phenotyping

#### Genotype

#### **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest.

# Representation of Amino Acid Changes

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' |
| | (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

A mutation as treatment emergent in class XX, the subject must have received a drug YY in class XX as part of their study treatment, and the mutation must be associated with resistance to a drug in class XX and not present at baseline.

#### **Resistance Associated Mutations**

• Known INI mutations associated with the development of resistance to RAL, EVG or DTG:

| Amino Acids in | H51Y, <b>T66A/I/K</b> , L74M, <b>E92Q/V</b> /G, Q95K, T97A, G118R, F121Y, E138A/K/D, |
|---|---|
| HIV Integrase for | G140A/C/S, <b>Y143C/H/R/K/S/G/A, P145S</b> , <b>Q146P</b> , <b>S147G</b> , <b>Q148H/K/R</b> , |
| Analysis | V151I/L/A, S153F/Y, N155H/S/T, E157Q, G163R/K, S230R, R263K, |
| | L68V/I*, L74I*, E138T*, V151I*, G193E* |

#### NOTES:

- Draft listing; may be modified in case of additional substantive data availability.
- INI mutations listed taken from Stanford HIV Resistance Database (http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI cited 28 Feb 2014) and accessed on 16 Feb 2015.
- Each INI mutation listed had a score of ≥15. INI substitutions listed above in bold had a score of =60.
- \* Denotes additional INI mutations added as they were identified during in vitro passage of DTG or seen in a

#### Genotype

#### **Amino Acid Changes**

previous DTG study in INI-experienced subjects (ING112574).

 Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis.

| Mutations |
|-------------------------------------------------------------------------|
| M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, |
| F116Y,<br>Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| D30N,V32I , M46I/L, I47A/V, G48V, I50V/L, I54M/L, Q58E, T74P, L76V, |
| V82A/T/F/L/S, N83D, I84V, N88S,L90M |

Note: List generated from IAS\_USA Guideline, [Wensing, 2014]

#### **Phenotype**

#### Phenotypic Susceptibility

- Phenotypic susceptibility to all licensed antiretroviral drugs and DTG will be determined using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change (FC) in IC50 relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.
- Since the maximum assay limit for FC for each ART varies from subject to subject, FC values
  that are greater than the maximum assay limit (e.g., '>100') will be interpreted as having a value
  equal to the smallest maximum assay limit for that ART in the study population for data
  analysis. Censored values will be presented 'as is' in the listings.
- Phenotypic susceptibilities will be categorised according to FC (based on Monogram PhenoSense assay). Clinical cut-offs (where available) or biological cut-offs by PhenoSense will be used to define the phenotypic susceptibility of background treatment.
- Replication capacity is generated as part of standard phenotypic assays.

| Drug | Abbreviation | Class | PhenoSense cutoff |
|---------------|--------------|-------|--------------------------|
| Abacavir | ABC | NRTI | (4.5 – 6.5) <sup>a</sup> |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |

| Phenotype | | | |
|---|---|---|---|
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivarine | RPV | NNRTI | 2 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| a. clinical cutoff (lower | cutoff – higher cutoff) | <u>.</u> | |

#### 12.6.6. Health outcomes

#### **HIVTSQs**

#### **Treatment Satisfaction Total Score**

- Items 1 to 10 are summed to produce a score with a possible range of 0 to 60.
- Higher scores represent greater treatment satisfaction as compared to the past few weeks.
- A maximum of 5 items can be missing, which can be imputed to reflect the mean of the completed item scores. If 6 or more items are missing, then the overall treatment satisfaction scale score should not be computed and will remain missing.

#### General Satisfaction/Clinical Sub-Score

- Items 1, 2, 3, 9, and 10 are summed to produce a score with a possible range of 0 to 30.
- Higher scores represent greater treatment satisfaction within this subscale as compared to the past few weeks.
- These subscales can be computed if at least 4 out of 5 items are available, in which case, the
  missing item can be imputed to reflect the mean of the completed item scores. If 2 or more
  items are missing, the score should not be computed and remain missing.

#### Lifestyle/Ease Sub-Score

- Items 4, 5, 6, 7, and 8 are summed to produce a score with a possible range of 0 to 30.
- Higher scores represent greater treatment satisfaction within this subscale as compared to the past few weeks.
- These subscales can be computed if at least 4 out of 5 items are available, in which case, the
  missing item can be imputed to reflect the mean of the completed item scores. If 2 or more
  items are missing, the score should not be computed and remain missing.

#### Individual Item Scores

Items are rated as 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied,

inconvenient, inflexible, etc.).

- Higher scores represent greater satisfaction with each aspect of treatment.
- Missing scores will not be computed and should remain missing.

# SF-12

# Physical Component Score (PCS) and Mental Component Score (MCS)

• Scores are created according to the manual [Ware, 1996] and are scored using software purchased from Quality Metric http://www.qualitymetric.com/.

# 12.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| <b>Element</b> General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as: <ul> <li>Randomized to ATV+RTV+TDF/FTC FDC and completed the Randomized Phase including the Week 48 Study Visit;</li> <li>Randomized to DTG/ABC/3TC FDC, completed the Randomized Phase including the Week 48 Visit, and did not enter the Continuation Phase;</li> <li>Randomized to DTG/ABC/3TC FDC, completed the Randomized Phase, including the Week 48 study visit, entered and completed the Continuation Phase (defined as remaining on study until commercial supplies of DTG/ABC/3TC become locally available or development of DTG/ABC/3TC is terminated).</li> </ul> </li> </ul> |
| | Withdrawn subjects were not replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed. |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| | <ul> <li>Unless stated, no imputation for missing data or premature discontinuation will<br/>be performed and the observed values will be used.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Health<br>Outcomes<br>HIV TSQ | For the HIV Treatment Satisfaction overall score (which is comprised of all 10 items), a maximum of 5 items may be missed and each computed as the mean of the completed item scores (as discussed in [Woodcock, 2006; Woodcock, 2001] |
| | <ul> <li>If 6 or more items are missed, then the overall score should not be<br/>computed and instead be imputed using LOCF.</li> </ul> |
| | <ul> <li>For the lifestyle/ease sub-score (which is comprised of 5 items), a maximum of 1 item may be missed and computed as the mean of the completed item scores.</li> <li>If 2 or more items are missed, then the overall score should not be computed and instead be imputed using LOCF.</li> </ul> |
| | For the convenience item and other individual item scores, missing scores will not be computed (according to Page 7 of the [HIVTSQ User Guidelines]) and |

| Element | Reporting Detail |
|---------|--------------------------------|
| | instead be imputed using LOCF. |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Exposure | If study treatment stop date is missing, then for the purposes of calculating exposure, it will be imputed using the date of last visit or the recorded date of withdrawal/completion whichever is earlier. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing.</li> <li>Any partial dates for adverse events will be raised to data management.</li> </ul> |
| | <ul> <li>If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month, unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases.</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> </ul> |
| | For medications recorded in the eCRF as prior ART, the earlier of this imputed date or the day before IP start will be used. The recorded partial date will be displayed in listings. |

#### 12.7.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Snapshot | <ul> <li>In the Snapshot dataset, subjects without HIV-1 RNA data in the assessment window for the visit of interest (due to missing data or discontinuation of IP prior to the visit window) are classified as non-responders in the derivation of the proportion of subjects with HIV-1 RNA &lt; 50 c/mL (or &lt;400 c/mL). The nature of this missing data will be further classified in Snapshot summaries as either 'Virologic Failure' or 'No Virologic Data at Week X'; see Section 12.11 for full details</li> </ul> |
| LOCF | In the LOCF dataset, missing values will be carried forward from the previous, non-missing available on-treatment assessment. |
| Lipid LOCF | <ul> <li>If subjects initiate serum lipid-lowering agents Post-baseline, then the last available fasted On-treatment lipid values prior to the initiation will be used in place of future, observed On-treatment values.</li> <li>Imputation will continue even if the subject discontinues the lipid-lowering agent.</li> <li>Missing assessments will not be imputed. Subjects on lipid-lowering agents at baseline will be excluded from this dataset.</li> </ul> |
| | This dataset will be used for all summaries of lipids data. |

# 12.8. Appendix 8: Values of Potential Clinical Importance

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values and | The DAIDS grading for severity of laboratory toxicities and clinical adverse events is included in the protocol. |
| Adverse<br>Events | The central laboratory will flag lab parameter toxicities directly in the provided datasets. |
| ECG | QTc above 500 msec or change from baseline above 60 msec are considered to be values of potential clinical importance. |

# 12.9. Appendix 9: Examination of Covariates and Subgroups

# 12.9.1. Handling of Covariates, Subgroups & Other Strata

- The following is a list of covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses (See Section 9.1.1 for further details).
- Additional covariates of clinical interest may also be considered.
- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Category | Covariates and / or Subgroups |
|---|---|
| Randomisation Strata | Randomisation is stratified by screening plasma HIV-1 RNA and CD4+ cell count, although summaries and analyses will make use of the Baseline categories, which are considered to be more relevant to the analysis of the study endpoints: ■ Baseline plasma HIV-1 RNA (≤ vs. >100,000 c/mL) ■ Baseline CD4+ cell count (≤ vs. >350 cells/mm³). All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| Demographic and Baseline<br>Characteristic Subgroups | <ul> <li>Age: ≥50 &amp; &lt;50</li> <li>Race: <ul> <li>White; Non-White</li> <li>African American/African Heritage; Non-African American/African Heritage</li> </ul> </li> <li>Country <ul> <li>Baseline plasma HIV-1 RNA: <ul> <li><li>&lt;1000; 1000 to &lt;10,000; 10,000 to &lt;50,000; 50,000 to 100,000; &gt;100,000 c/mL.</li> <li>Baseline CD4+ cell count: <ul> <li>&lt;50; 50 to &lt;200; 200 to &lt;350; 350 to &lt;500; ≥500 cells/mm3.</li> <li>Baseline Centers for Disease Control and Prevention (CDC) category:</li></ul></li></li></ul></li></ul></li></ul> |

# 12.10. Appendix 10: Model Checking and Diagnostics for Statistical Analyses

#### 12.10.1. Statistical Analysis Assumptions

| Endpoint(s) | Change from Baseline in fasted lipids (triglycerides and TC/HDL ratio) |
|---|---|
| Analysis | Multiple imputation |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals (i.e. checking the normality assumption) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.
- Diagnostic plots (trace and autocorrelation plots) will be checked to verify that the number of burn-in iterations and MCMC steps between imputed datasets are sufficient. If the trace plots show apparent trend or the autocorrelation plots show significant positive or negative autocorrelation, number of iterations will be increased until the diagnostic plots are acceptable.

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be estimated by treatment group by specifying 'type=UN' and 'group=treat' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

## 12.11. Appendix 11: Snapshot

#### **Detailed Algorithm Steps**

- Consider an arbitrary visit window, Week X (see Section 12.3).
- A subject's response (i.e., 'Virologic Success', 'Virologic Failure', or 'No Virologic Data at Week X') in that window is determined as indicated below, in the order stated.
- If non-permitted change in background ART prior to Week X: <u>Subject = Virologic Failure</u>.
- If permitted change in background ART prior to Week X AND decision to make this change is after the first On-treatment HIV-1 RNA result AND the latest On-treatment HIV-1 RNA result prior to the date of decision to switch is ≥ 50 c/mL: Subject = Virologic Failure.
- 3. If non-permitted change in background ART during Week X

OR

if permitted change in background ART **during** Week X AND decision to make this change is *after* the first On-treatment HIV-1 RNA result AND the latest On-treatment HIV-1 RNA result prior to the date of decision to switch is >=50 c/mL

#### AND:

- no HIV-1 RNA result is available during Week X prior to change: <u>Subject = Virologic Failure</u>;
- there is at least one HIV-1 RNA result available during Week X prior to the change, then consider the latest such result:
  - If < 50 c/mL: <u>Subject = Virologic Success</u>
  - If ≥ 50 c/mL: Subject = Virologic Failure.
- 4. If there is no change in background ART prior or during Week X

OR

a permitted change **prior or during** Week X is decided on *before* the first On-treatment HIV-1 RNA result,

OR

a permitted change **prior or during** Week X is decided on *after* the first On-treatment RNA result AND the latest On-treatment HIV-1 RNA result prior to the decision to switch is <50 c/mL,

AND

at least one HIV-1 RNA result is available during Week X, then consider the latest such result:

- If < 50 c/mL: Subject = Virologic Success:</li>
- If ≥ 50 c/mL: Subject = Virologic Failure.
- If there is no change in background ART prior or during Week X

OR

a permitted change **prior or during** Week X is decided on *before* the first On-treatment HIV-1 RNA result

#### **Detailed Algorithm Steps**

OR

a permitted change **prior or during** Week X is decided on *after* the first On-treatment RNA result AND the latest On-treatment HIV-1 RNA result prior to the decision to switch is <50 c/mL,

#### AND

no HIV-1 RNA results are available during Week X:

- If the subject has not withdrawn from the study prior to or during Week X: <u>Subject = No Virologic Data at Week X</u>, with a reason of 'Missing data during window but on study';
- If the subject was withdrawn from the study prior to or during Week X due to AE or death: <u>Subject = No Virologic Data at Week X</u>, with a reason of 'Discontinued due to AE or Death':
- Otherwise, consider the subject's last available On-treatment HIV-1 RNA result:
  - ➤ If <50 c/mL or no result is available: <u>Subject = No Virologic Data at Week X</u>, with a reason of 'Discontinued for Other Reasons';
  - If ≥ 50 c/mL: Subject = Virologic Failure.

#### **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

• HIV-RNA = 580 copies/mL at Day 336, HIV-RNA below 50 copies/mL on Day 350. This should be categorized as Virologic Success.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be
  classified as Discontinued due to AE or Death (as appropriate), regardless of the HIV-RNA
  result, even if the HIV-RNA is below 50 copies/mL at the time of discontinuation.
- However, if a patient has an HIV-RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response. This is the Virology First hierarchy:
  - a. HIV-RNA below 50 copies/mL at Day 336 and discontinues because of AE or even dies on Day 360 this person is categorized as <u>Virologic Success</u>.
  - b. HIV-RNA is 552 copies/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as Virologic Failure.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as Discontinued for Other Reasons.
- If a patient discontinues the study before the window because of *lack of efficacy* then the patient should be included in the <u>Virologic Failure</u> row and not in the <u>Discontinued</u> for

#### **Detailed Algorithm Steps**

Other Reasons row.

- If a patient discontinues because of subject withdrew consent and his or her HIV-1 RNA
  result at the time of discontinuation was equal to or above 50 copies/mL, then he or she
  should be categorized as Virologic Failure and NOT as Discontinued for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-RNA result was 49 copies/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment *not permitted by protocol* they should be considered an efficacy failure and captured as <u>Virologic Failure</u>.

#### On study but missing data in window:

- If there are no data during Days 295 to 378, but there is an HIV-RNA below 50 copies/mL on Day 380, this patient should be considered *On Study but Missing Data in Window.*
- If there are no data during Days 295 to 378, but there is an HIV-RNA equal to or above 50 copies/mL on Day 280, this patient also should be classified as On Study but Missing Data in Window.

#### Optimized Background Therapy Substitutions After Randomization

 OBT substitutions (in-class or cross-class) permitted per protocol for documented toxicity reasons can be permitted on or before the first trial visit without penalty.

If OBT substitutions for toxicity reasons occur after the first trial visit, then patients should be categorized as <u>Virologic Failure</u> if they have HIV-RNA above 50 copies/mL at the time of switch.

# 12.12. Appendix 12: Abbreviations & Trade Marks

# 12.12.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ABC | Abacavir |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ALT | Alanine aminotransferase |
| ART | Antiretroviral Treatment |
| ATC | Anatomical Therapeutic Chemical |
| ATV | Atazanavir |
| c/ml | Copies per milliliter |
| CDC | Centers for Disease Control and Prevention |
| CDISC | Clinical Data Interchange Standards Consortium |
| CD4+ | Helper-inducer T-lymphocyte having surface antigen CD4 (cluster of |
| | differentiation 4) |
| CI | Confidence Interval |
| CMH | Cochran-Mantel-Haenszel |
| CRT | Serum creatinine |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CV | Cardiovascular |
| DAIDS | Division of AIDS |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| ERDF | Efficacy Related Discontinuation = Failure |
| FC | Fold change |
| FDA | Food and Drug Agency |
| FDC | Fixed Dose Combination |
| FU | Follow-up |
| GFR | Glomerular Filtration Rate |
| GSK | GlaxoSmithKline |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HDL | High density lipoprotein |
| HIV(-1) | Human immunodeficiency virus (type 1) |
| HIVTSQs | HIV Treatment Satisfaction Questionnaire |
| HSR | Hypersensitivity reaction |
| IAS-USA | International Antiviral Society-USA |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IG | Implementation Guide |
| IN(I) | Integrase (Inhibitor) |
| IP | Investigational Product |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| ITT(E) | Intent-To-Treat (Exposed) |
| LDL | Low density lipoprotein |
| LOCF | Last Observation Carries Forward |
| LVH | left ventricular hypertrophy |
| MAR | Missing at random |
| MCMC | Markov Chain Monte Carlo |
| MCS | Mental Component Score |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| MMRM | Mixed Model Repeated Measures |
| NCEP | National Cholesterol Education Program |
| NNRTI | Non-nucleoside Reverse Transcript Inhibitor |
| NRTI | Nucleoside Reverse Transcript Inhibitor |
| OC | Observed Case |
| PCS | Physical Component Score |
| PDMP | Protocol Deviation Management Plan |
| PI | Protease Inhibitor |
| PP | Per Protocol |
| PSRAE | Possibly suicidality related Adverse Event |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RNA | Ribonucleic acid |
| RTF | Rich text format |
| RTV | Ritonavir |
| RUCAM | Roussel Uclaf Causality Assessment Method |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Software |
| SBP | Systolic blood pressure |
| SDTM | Study Data Tabulation Model |
| SF-12 | 12-Item Short Form |
| SOC | System Organ Class |
| TC | Total Cholesterol |
| TDF/FTC | Tenofovir/emtricitabine |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation = Failure |
| VF | Virologic Failure |

#### 12.12.2. Trademarks

| Trademarks of ViiV Healthcare |
|-------------------------------|
| Dolutegravir |
| Epzicom/Kivexa |

| Trademarks not owned by ViiV<br>Healthcare |
|--------------------------------------------|
| Norvir |
| Reyataz |
| SAS |
| Truvada |
| TSCG |
| TYLENOL |

# 12.13. Appendix 13: Final (End of Study) Analysis

This appendix provides the details of the planned analyses and data displays for ING117172 End of Study (EoS) reporting.

The primary analysis (i.e. interim analysis at Week 48) was completed based on the original RAP. This appendix is written to cover only analyses included in the final end of study reporting. All derivations described in the study analysis plan will be re-used for end of study reporting and only those definitions and derivations that have changed since the previous interim analysis are described below. This additional appendix summarizes only the key endpoints of interest for the final analysis and explain any deviations from the primary analysis. The details of the final EOS reporting and analysis plan are described below:

- 1. The analysis for which the data have not been changed since last interim analysis will not be reported to avoid redundancy. These reports include the analyses of demographic and baseline characteristics.
- 2. No subgroup analysis, hypotheses testing, or statistical analyses will be performed.
- 3. All required disclosure outputs following the FDAAA and EudraCT guidelines will be produced.
- 4. For the purpose of creation of Mexico Final Safety Report and submission to Ministry of Health, some listings at Mexico sites will be reported separately. Such listings are identified in the Programming notes in Section 12.13.8. These listings will include data from both Randomized and Continuation Phase.
- 5. All by visit tables will have all visits reported from both Randomized and Continuation Phase.
- 6. All listings that include both Randomized and Continuation Phase data will have the Phase mentioned in the outputs except for Listing of Investigational Product Exposure Data.

#### 12.13.1. Study Phases

In previous analysis (primary Week 48 reporting), data were summarized only for the Randomized phase of the study. However, when data from the Continuation phase were available, certain displays were repeated for the combined time period of Randomized plus Continuation phases. For EoS reporting, if for any display, data from both study phases (Randomized phase plus Continuation phase) are included, they will be tabulated in one summary table, unless specified otherwise, and it will be noted in the title of the output. For listings that contain all the data, a new column will be added to specify the phase of the study for each record.

Start and end date for Randomized and open-label phases are defined as follows:

| Study Treatment Date | <u>Definition</u> |
|---|---|
| Randomized phase treatment start date | The earliest exposure start date, where investigational product is either DTG/ABC/3TC or ATV+RTV+TDF/FTC |
| Randomized phase treatment end date | <ul> <li>If Treatment arm= ATV+RTV+TDF/FTC</li> <li>Randomized phase treatment end date= Last non-missing exposure date.</li> <li>If Treatment arm= DTG/ABC/3TC</li> <li>Randomized phase treatment end date= Week 48 visit date or unscheduled Week 48 visit date.</li> <li>If the participant discontinued the study before Week 48, then Randomized phase treatment end date= Last non-missing exposure end date</li> </ul> |
| Continuation phase treatment start date | <ul> <li>Randomization phase treatment end date+1 day where Treatment arm = DTG/ABC/3TC</li> <li>There will be no Continuation phase if Treatment arm= ATV+RTV+TDF/FTC.</li> </ul> |
| Continuation phase treatment end date | The last non-missing exposure end date after<br>entering the Continuation Phase in the<br>DTG/ABC/3TC arm. |

# 12.13.1.1. Study Phases for all events that do not have visits associated with them

| Phase | Definition |
|---|---|
| | Randomized phase treatment start date ≤ Event Start Date ≤Randomized phase end date |
| Continuation Phase Event | Event Start Date ≥ Continuation phase treatment start date |

Note: In the case of a completely missing start date, the event will be considered to have started in the Randomized Phase.

#### 12.13.1.2. Treatment Phases for Concomitant/Post-Therapy Medications Data

- For subjects who do not enter into Continuation phase, all <u>on-treatment and post-treatment</u> concomitant medications (conmeds) will be in Randomized phase;
- For subjects who enter into Continuation phase; all <u>on-treatment and post-treatment</u> conmeds will be in Randomized phase, Continuation phase or both (Randomized + Continuation) phases depending on the conmeds start/stop dates.
  - o Randomized phase- If the conmeds end dates < Continuation treatment start date.
  - Continuation phase- If the conmeds start dates ≥Continuation treatment start date.
  - o Randomized and Continuation-
    - If conmed start date
       Continuation treatment start date + conmed end date
       Continuation treatment start date
    - If conmed start date
       Continuation treatment start date + conmed end date= missing
    - If conmed start date= missing + conmed end date≥ Continuation treatment start date
    - If conmed start date= missing + conmed end date= missing

# 12.13.2. Analysis Populations for the Continuation Phase

The following populations have been defined only for the Continuation Phase. For all other populations refer to Section 5.

| Population | Definition/ Criteria. | Analysis Evaluated |
|---|---|---|
| Safety- Continuation Phase | Comprises of all subjects in<br>the DTG/ABC/3TC arm who<br>receive at least one dose of<br>study treatment after entering<br>the Continuation Phase. | |

| Population | Definition/ Criteria. | Analysis Evaluated |
|---|---|---|
| | Comprises of all subjects in<br>the ITT-E population (as<br>defined in Section 5) in the<br>DTG/ABC/3TC arm who<br>enter the Continuation Phase | Study Population |

### 12.13.3. Study Population

The study population summaries and data listings will be based on the ITT-E or ITT-E-Continuation Phase population, unless otherwise specified. Subject accountability summary will be produced for the overall study and separately for the Continuation Phase. Overview of the key planned study population endpoints:

- Study Populations
- Subject Accountability
- Concomitant and Antiretroviral Medications
- Protocol deviations

#### 12.13.4. Safety Analysis

All safety displays will be based on the Safety population or Safety-Continuation Phase Population. The core adverse event displays for the final report have been identified based on the IDSL library required tables. For AE data (including COVID-19), unless stated otherwise, the summaries and listings will include only those AEs that occurred during Continuation Phase.

Summaries of AE required for the FDAAA and EudraCT will be generated in this reporting effort. Such summaries are identified in the Programming notes. These summaries will include participants from both Randomized and Continuation Phase. Common AEs are those with >=3% (without rounding) incidence for any treatment. One figure will be reported to present Maximum ALT vs. Maximum Total Bilirubin. Overview of the key planned safety endpoints:

- Extent of Exposure
- Adverse Events
- Maximum Post-Baseline Emergent Clinical Chemistry/ Haematology Toxicities/ Hepatobiliary Laboratory Abnormality Criteria
- Liver Events Assessment
- Positive Suicidal indication Alerts based on eC-SSRS will be listed including data only in the Continuation Phase
- For subjects at Mexico sites and non-Mexico sites the following listings will be generated in this reporting effort. These listings will include data from both Randomized and Continuation Phase.
  - Listing of Non-Serious AEs of Subjects at Mexico sites
  - Listing of SAEs of Subjects at Mexico sites

Listing of SAEs of Subjects at non-Mexico sites

# 12.13.5. Efficacy Analysis

The efficacy summaries and data listings will be based on the ITT-E population, unless otherwise specified. Subjects Randomized to the ATV+RTV+TDF/FTC arm completed the study after the Week 48 visit. Thus, the Snapshot algorithm that was used in the previous interim analyses would not be appropriate. Instead, HIV-1 RNA viral load will be summarized using observed data (i.e., subjects with missing data at a time point are excluded). The summaries and listings will be based on both Randomized and Continuation phase. Overview of the key planned efficacy endpoints:

- Absolute values in Plasma HIV-1 RNA and CD4+ Cell counts over time
- Proportion of Subjects with Plasma HIV-1 RNA < 50 c/ mL- observed data
- Proportion of subjects with Confirmed Virologic Withdrawal based on observed data.
- Change from Baseline in CD4+ cell count (cells/mm3) and Plasma HIV-1 RNA (log10 c/mL) by Visit
- Incidence of disease progression and HIV- associated conditions

#### 12.13.6. Virology Analysis

The Virology displays will be based on ITT-E or Viral Genotypic and Viral Phenotypic populations. All virology summaries and Listings will include subjects who met Confirmed Virologic Withdrawal criteria during both Randomized and Continuation phase by separating the phases by page. Resistance testing will be performed on subjects at non-CVW time (ie, last on-treatment VL>400), and these subjects' viral data will be included only in the listing of resistance data for subjects at non-CVW time.

Prespecified lists of integrase substitutions have been modified since the previous interim analysis, hence an updated list of known INSTI mutations has been added in Table 8 and IAS-USA major resistance associated mutations (RAMs) to other classes (i.e., NRTI, NNRTI, PI) are listed in Table 9.

#### 12.13.6.1. Genotype

# Table 8 Known INSTI mutations associated with the development of resistance to RAL, EVG or DTG

| Amino Acids | H51Y, <u><b>T66A/I/K</b></u> , L74M, <u><b>E92Q/V</b>/G</u> , Q95K, T97A, G118R, <u><b>F121Y</b></u> , E138A/K, |
|---|---|
| in HIV | G140A/C/S, <u>Y143C/H/R/K/S/G/A</u> , <u>P145S</u> , <u>Q146P</u> , <u>S147G</u> , <u>Q148</u> N/ <u>H/K/R</u> , |
| Integrase for | <b>V151</b> I/L/A, S153F/Y, <b>N155</b> H/S/T, E157Q, G163R/K, S230R, R263K, |
| Analysis | L68V/I*, L74I*, E138T*, G193E* |

#### **NOTES:**

- Current listing includes INSTI mutations identified via the Stanford HIV Resistance database, or identified during in vitro passage of DTG, or as seen in a previous DTG studies in INSTIexperienced subjects (i.e. ING112574) and may be modified in case of additional substantive data availability.
- INSTI mutations in bold have the maximum score of 60 and are for any INSTI drug in the Stanford database v8.9 (http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INSTI last updated on 25 OCT 2019 and accessed on 17 FEB 2020); the rest have a maximum score <60.
- The INSTI mutations listed are historically identified via the Stanford HIV Resistance database, and also include mutations identified during in vitro passage of DTG, or as seen in a previous DTG study in INSTI-experienced subjects (ING112574).

Table 9 Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA).

| Class | Mutations |
|---|---|
| NRTIs | M41L, K65R/E/N, D67N, 69 insert, K70E/R, L74V, Y115F, M184V/I, L210W, T215Y/F, K219Q/E; [A62V, V75I, F77L, F116Y, Q151M] |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138A/G/K/Q/R, V179L,Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L |
| PIs | D30N,V32I , M46I/L, I47A/V, G48V, I50V/L, I54V/M/L, Q58E, T74P, L76V, V82A/T/F/L/S, N83D, I84V, N88S, L90M |

#### NOTES:

- Updated to "2019 Resistance Mutations Update Volume 27 Issue 3, July/August 2019
- The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis.
- Q151M Complex: Q151M usually occurs in combination with two or more of the following four accessory NRTI mutations A62V, V75I, F77L, and F116Y. However, if any one of these mutations occur alone, they shall be considered as major mutation for the NRTI class.

A mutation as treatment emergent in class XX, the subject must have received a drug YY in class XX as part of their study treatment, and the mutation must be associated with resistance to a drug in class XX and not present at baseline.

### Stanford Genotypic Susceptibility Score (GSS)

- To establish genotypic susceptibility to ART treatment, a genotypic sensitivity score will be calculated.
- Genotypic sensitivity to each drug will be assessed using the HIVdb, the Integrated Genotypic Resistance Interpretation System [Liu, 2006].
- In the HIVdb system, each HIV-1 drug resistance mutation is assigned a drug penalty score. The penalty scores for each drug resistance mutation are available at

NNRTI: https://hivdb.stanford.edu/dr-summary/mut-scores/NNRTI/

NRTI: https://hivdb.stanford.edu/dr-summary/mut-scores/NRTI/

PI: https://hivdb.stanford.edu/dr-summary/mut-scores/PI/

INSTI: <a href="https://hivdb.stanford.edu/dr-summary/mut-scores/INSTI/">https://hivdb.stanford.edu/dr-summary/mut-scores/INSTI/</a>. Scores for particular patterns of INSTIs are also available at <a href="https://hivdb.stanford.edu/dr-summary/pattern-scores/INSTI/">https://hivdb.stanford.edu/dr-summary/pattern-scores/INSTI/</a>.

The drug resistance estimate is obtained by adding together the penalty scores from all mutations associated with resistance to that drug and then a numeric score (GSS) is applied for each drug as shown below. The sum scores are titrated to fall within the following ranges susceptible, potential low-level resistance, low-level resistance, intermediate resistance, and high-level resistance (see table below).

| Resistance<br>Estimate | S-GSS Score | Sensitivity |
|------------------------|-------------|--------------------------------|
| 0 – 9 | 1 | Susceptible |
| 10 – 14 | 0.75 | Potential low-level resistance |
| 15 – 29 | 0.5 | Low-level resistance |
| 30 – 59 | 0.25 | Intermediate resistance |
| ≥60 | 0 | High-level resistance |

The HIVdb GSS will then be calculated for each subject defined as the sum of the resistance scores for each component of their drugs.

#### 12.13.6.2. Phenotype

To establish susceptibility to background treatment, a phenotypic sensitivity score will be calculated. Phenotypic susceptibility to each drug in a subject's background regimen will be determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold resistance to that drug at a certain timepoint (e.g., Screening or Baseline). A numeric score will be assigned to each background drug using two different methods: one with full sensitivity only (PSSf) and one with partial sensitivity included (PSSp).

# PSS with Full Sensitivity Only (PSSf)

| Fold Change | Score | Interpretation |
|--------------------------------------------|-------|----------------|
| > clinical lower cutoff or biologic cutoff | 0 | resistance |
| ≤ clinical lower cutoff or biologic cutoff | 1 | sensitive |

# PSS with Partial Sensitivity Included (PSSp)

| Fold Change | Score | Interpretation |
|---|---|---|
| > clinical higher cutoff | 0 | resistance |
| ≤ clinical higher cutoff and > clinical lower cutoff | 0.5 | partially sensitive |
| ≤ clinical lower cutoff | 1 | sensitive |

Both PSSf and PSSp will be calculated separately for each subject defined as the sum of the resistance scores for each background drug.

Clinical and Biological Cutoff Values for the PhenoSense HIV Drug Resistance Assay have changed since the previous interim analysis, hence for EoS phenotypic susceptibility will be categorised according to Fold Change as shown in Table 10 (based on Monogram PhenoSense assay).

Table 10 Clinical and Biological Cutoff Values for the PhenoSense HIV Drug Resistance Assay

| Drug | Abbreviation | Class | PhenoSense Cutoff |
|-----------------|--------------|-------|-----------------------|
| Abacavir | ABC | NRTI | $(4.5-6.5)^a$ |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddI | NRTI | $(1.3-2.2)^a$ |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) <sup>a</sup> |
| Rilpivirine | RPV | NNRTI | 2.5 |
| Fosamprenavir | FPV | PI | 2 a,c |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir | ATV | PI | 2.2 a, |
| Atazanavir/r | ATV/r | PI | 5.2 a,c |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | $(9-55)^{a}$ |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir | SQV | PI | 1.7 a,c |
| Saquinavir/r | SQV/r | PI | $(2.3-12)^{a}$ |
| Tipranavir/r | TPV/r | PI | $(2-8)^{a}$ |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 <sup>b</sup> |
| Raltegravir | RAL | INSTI | 1.5 |
| Elvitegravir | EVG | INSTI | 2.5 |
| Dolutegravir | DTG | INSTI | (4-13) a |

a: clinical cutoff (lower cutoff – higher cutoff)

Overview of the key planned virology endpoints:

- Genotypic and Phenotypic Accountability
- Major Mutations in NNRTI, NRTI and PI Classes and Pre-specified Mutations in INSTI from Baseline to Time of CVW
- Fold Change Summary of Fold Change to DTG at Baseline and Time of CVW

b: standard cut-off used by Monogram Inc. until clinical or biological cutoff have been determined

c: Only the boosted cutoff shall be used to compute the PhenoSense sensitivity for Atazanavir,

Fosamprenavir and Saquinavir except stated otherwise.

# 12.13.7. COVID-19 Analysis

This study started in 2013 and is being continued during the outbreak of the ongoing COVID -19 pandemic. The information regarding the number of subjects affected by COVID-19 and its symptoms will be reported according to GSK core standards. The visits impacted due to the pandemic outbreak will be reported. Protocol deviations or adverse events related to COVID-19 if any, will also be reported according to GSK core standards.

## 12.13.8. List of Data Displays for Final (End of Study)

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 1.1 | All<br>Subjects<br>Screened | SA1 | Summary of Study Populations | CS CORE;<br>Only add the<br>populations that<br>will be used for<br>EOS | EOS |
| 1.7 | ITT(E) -<br>Continuation<br>Phase | DV1a | Summary of Important Protocol<br>Deviations by relationship to<br>COVID-19 Pandemic-<br>Continuation Phase | CS CORE | EOS |

| Study Population Tables | | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable | | |
| 1.27 | ITT(E) -<br>Continuation<br>Phase | Same as<br>Week 48<br>Table<br>1.27 | Summary of Subjects by Country and Investigator- Continuation Phase | | EOS | | |
| 1.28 | ITT(E) | ES1 | Summary of Subject Status and<br>Subject Disposition by<br>Relationship to COVID-19<br>Pandemic | FDAAA, EudraCT For overall, both phases Summarise by: i) Overall ii) Related to COVID-19, ii) Not related to COVID-19 | EOS | | |
| 1.29 | ITT(E) -<br>Continuation<br>Phase | ES1 | Summary of Subject Status and<br>Subject Disposition by<br>relationship to COVID-19<br>Pandemic- Continuation Phase | New Output; FDAAA, EudraCT Summarise by: i) Overall ii) Related to COVID-19, ii) Not related to COVID-19 | EOS | | |
| Effica | Efficacy Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming Notes | Deliverable | | | |
| 2.7 | ITT(E) | Same shell as ARIA Week<br>48 Table 2.7 | Summary of Change<br>from Baseline in<br>Plasma HIV-1 RNA<br>(log10 c/mL) by Visit | | EOS | | | |
| 2.13 | ITT(E) | Same shell as ARIA Week<br>48 Table 2.13 | Proportion of Subjects Meeting Confirmed Virologic Withdrawal Criteria by Visit- Observed Case | | EOS | | | |
| 2.15 | ITT(E) | Same shell as ARIA Week<br>48 Table 2.15 | Summary of Change<br>from Baseline in CD4+<br>Cell Count<br>(cells/mm^3) by Visit | | EOS | | | |
| 2.16 | ITT(E) | HIV1 | Summary of Post-<br>Baseline HIV-1<br>Associated Conditions<br>Including Recurrences | | EOS | | | |
| 2.17 | ITT(E) | HIV1 | Summary of Post-<br>Baseline HIV-1<br>Associated Conditions<br>Excluding<br>Recurrences | | EOS | | | |
| 2.18 | ITT(E) | HIV2 | Summary of Post-<br>Baseline HIV-1<br>Disease Progressions | | EOS | | | |
| 2.19 | ITT(E) | gsk2619619/mid200336/<br>final_01/table 2.1 | Proportion of Subjects<br>with Plasma HIV-1<br>RNA <50 c/mL by Visit<br>– Observed Case | | EOS | | | |
| 2.20 | ITT(E) | gsk2619619/mid200336/<br>final_01/table 2.41 | Summary of Absolute values in plasma HIV-1 RNA over time | | EOS | | | |
| 2.21 | ITT(E) | gsk2619619/mid200336/<br>final_01/table 2.41 | Summary of CD4+ cell counts over time | | EOS | | | |

#### **CONFIDENTIAL**

ING117172

| Effica | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 2.4 | ITT(E) | Same<br>shell as<br>Gemini<br>Figure<br>2.3 | Individual Plasma HIV-1 RNA (log10 c/mL) and CD4+ Profiles by Visit for Subjects with at least One Suspected Virologic Withdrawal Visit | | EOS |

| Safety Ta | Safety Tables | | | | |
|---|---|---|---|---|---|
| No | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 3.2 | Safety | Same<br>shell as<br>Week 48<br>table 3.1 | Summary of Extent of<br>Exposure to Investigational<br>Product | CS Core | EOS |
| 3.52 | Safety-<br>Continuation<br>Phase | Same<br>shell as<br>Week 48<br>table 3.1 | Summary of Extent of<br>Exposure to Investigational<br>Product – Continuation Phase | New output | EOS |
| 3.3 | Safety-<br>Continuation<br>Phase | AE5 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity- Continuation Phase | CS Core | EOS |
| 3.4 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency- Continuation Phase | CS Core | EOS |
| 3.5 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Common (>=3%)<br>Grade 2-4 Adverse Events by<br>Overall Frequency-<br>Continuation Phase | CS Core | EOS |
| 3.6 | Safety-<br>Continuation<br>Phase | AE5 | Summary of All Drug-Related<br>Adverse Events by System<br>Organ Class and Maximum<br>Toxicity- Continuation Phase | CS Core | EOS |
| 3.7 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Common (>=3%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency- Continuation Phase | CS Core | EOS |
| 3.8 | Safety-<br>Continuation<br>Phase | AE16 | Summary of Serious Adverse<br>Events by System Organ<br>Class- Continuation Phase | | EOS |

| 3.9 | Safety | AE16 | Summary of Serious Adverse<br>Events by System Organ Class<br>and Preferred Term (Number<br>of Subjects and Occurrences) | CS Core New output. FDAAA, EudraCT | EOS |
|---|---|---|---|---|---|
| 3.11 | Safety-<br>Continuation<br>Phase | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product – Continuation Phase | CS Core | EOS |
| 3.13 | Safety | AE3 | Summary of Common (>=3%) Non-Serious Adverse Events | CS Core<br>FDAAA | EOS |
| 3.14 | Safety | AE15 | Summary of Common (>=3%) Non-Serious Adverse Events by System Organ Class and Preferred term (Number of Subjects and Occurrences) | CS Core<br>EudraCT | EOS |
| 3.29 | Safety-<br>Continuation<br>Phase | Same<br>shell as<br>Week 48<br>Table<br>3.29 | Summary of Maximum Post-<br>Baseline Emergent Chemistry<br>Toxicities –Continuation Phase | CS Core | EOS |
| 3.30 | Safety-<br>Continuation<br>Phase | Same<br>shell as<br>Week 48<br>Table<br>3.30 | Summary of Maximum Post-<br>Baseline Emergent<br>Hematology Toxicities –<br>Continuation Phase | CS Core | EOS |
| 3.41 | Safety-<br>Continuation<br>Phase | LIVER10 | Summary of Subjects Meeting Hepatobiliary Laboratory Abnormality Criteria Post- Baseline Emergent- Continuation Phase | | EOS |
| 3.42 | Safety-<br>Continuation<br>Phase | Same<br>shell as<br>ARIA<br>Week 48 | Subjects Meeting Hepatobiliary<br>Abnormality Criteria - Post-<br>Baseline Emergent-<br>Continuation Phase | | EOS |

#### **CONFIDENTIAL**

ING117172

| 3.50 | Safety-<br>Continuation<br>Phase | PAN1 | Summary of COVID-19 Assessment for Subjects with COVID-19 Adverse Events- Continuation Phase | New Output | EOS |
|---|---|---|---|---|---|
| 3.51 | Safety-<br>Continuation<br>Phase | PAN3 | Summary of COVID-19<br>Symptoms for Subjects with<br>COVID-19 Adverse Events-<br>Continuation Phase | New Output | EOS |

| Safety | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 3.3 | Safety-<br>Continuation<br>Phase | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin-Continuation Phase-Continuation Phase | CS CORE | EOS |
| 3.10 | Safety | gsk1349572/<br>ing111762/<br>final_01/<br>Figure 8.27 | Plot of cumulative exposure to Investigational Product | New output; | EOS |

| Virolo | Virology Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID / Example Shell | Title | Programmin g Notes | Deliverabl<br>e |
| 7.9 | Genotypic | PFG1 | Summary of Major Mutations in NNRTI, NRTI and PI Classes and Pre-specified Mutations in INSTI Class at Baseline and time of CVW for Subjects Meeting CVW Criteria | New Output; For EoS both phases will be included. | EOS |
| 7.1 | Genotypic | gsk1349572/mid200304/primary_0<br>1/ Table 12.1 | Summary of<br>Subject<br>Accountabilit<br>y: Genotypes<br>Available | New Output; For EoS both phases will be included. | EOS |
| 7.5 | Phenotypi<br>c | Same shell as Week 48 Table 7.5 | Summary of<br>Phenotype at<br>time of CVW<br>by<br>phenotypic<br>cut-off | For EoS<br>both phases<br>will be<br>included | EOS |
| 7.7 | Phenotypi<br>c | Same shell as Week 48 Table 7.7 | Summary of<br>Fold Change<br>at Baseline<br>and Time of<br>CVW | For EoS<br>both phases<br>will be<br>included. | EOS |
| 7.1<br>1 | Phenotypi<br>c | gsk1349572/mid200304/primary_0<br>1/ Table 12.6 | Summary of<br>Subject<br>Accountabilit<br>y:<br>Phenotypes<br>Available | New Output; For EoS both phases will be included. | EOS |

| ICH | ICH Listings | | | | |
|---|---|---|---|---|---|
| No | Populatio<br>n | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming Notes | Deliverabl<br>e |
| 4 | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | CS CORE | EOS |
| 6 | ITT-E-<br>Continuatio<br>n Phase | DV2 | Listing of Important<br>Protocol Deviations -<br>Continuation Phase | CS CORE | EOS |
| 79 | ITT-E-<br>Continuatio<br>n Phase | DV2 | Listing of All Non-<br>Important COVID-19<br>related Protocol<br>Deviations-<br>Continuation Phase | New Output | EOS |
| 10 | ITT-E | Same as<br>Week 48<br>listing 10 | Listing of<br>Quantitative Plasma<br>HIV-1 RNA Data | | EOS |
| 13 | Safety | HIV_IP<br>5 | Listing of Investigational Product Exposure Data | CS CORE | EOS |
| 16 | Safety-<br>Continuatio<br>n Phase | AE8 | Listing of All<br>Adverse Events-<br>Continuation Phase | CS CORE | EOS |
| 17 | Safety-<br>Continuatio<br>n Phase | AE8 | Listing of Fatal<br>Adverse Events-<br>Continuation Phase | CS CORE | EOS |
| 18 | Safety-<br>Continuatio<br>n Phase | AE8 | Listing of Non-Fatal<br>Serious Adverse<br>Events-Continuation<br>Phase | CS CORE | EOS |
| 19 | Safety-<br>Continuatio<br>n Phase | AE8 | Listing of Adverse Events Leading to Withdrawal/Permane nt Discontinuation of Investigational Product- Continuation Phase | CS CORE | EOS |

| ICH | ICH Listings | | | | |
|---|---|---|---|---|---|
| No | Populatio<br>n | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming Notes | Deliverabl<br>e |
| 20 | Safety-<br>Continuatio<br>n Phase | AE2 | Listing of Relationship of Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text- Continuation Phase | CS CORE | EOS |
| 22 | Safety | LB5 | Listing of Laboratory Data for Subjects with Grade 3 or 4 Post-Baseline Emergent Toxicities- Continuation Phase | Use the shell of Listing 56 from gsk1349572/mid200304/primary_ 01/ | EOS |
| 25 | Safety-<br>Continuatio<br>n Phase | PSRAE<br>1 | Listing of Possible Suicidality-Related Adverse Event Data: Event and Description (Section 1- Section 2) - Continuation Phase | | EOS |
| 26 | Safety-<br>Continuatio<br>n Phase | PSRAE<br>3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3)- Continuation Phase | | EOS |
| 27 | Safety-<br>Continuatio<br>n Phase | PSRAE<br>4 | Listing of Possible<br>Suicidality-Related<br>Adverse Event Data<br>(Section 4)-<br>Continuation Phase | | EOS |
| 28 | Safety-<br>Continuatio<br>n Phase | PSRAE<br>5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5- Section 8)- Continuation Phase | | EOS |

| Non- | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 29 | All<br>Subjects<br>Screened | Same shell as ARIA Week<br>48 Listing 29 | Listing of Study<br>Populations | | EOS |
| 32 | ITT-E | Same shell as ARIA Week<br>48 Listing 32 | Listing of Visit Dates | | EOS |
| 40 | ITT-E | Same shell as ARIA Week<br>48 Listing 40 | Listing of Investigational Product Accountability | | EOS |
| 41 | ITT-E-<br>Continuation<br>Phase | CM2 | Listing of Concomitant Medications- Continuation Phase | CS CORE | EOS |
| 45 | ITT-E-<br>Continuation<br>Phase | CM2 | Listing of Concomitant ART Medications- Continuation Phase | | EOS |
| 48 | ITT-E | Same shell as ARIA Week<br>48 Listing 48 | Listing of Subjects with Confirmed Virologic Withdrawal | Data in both<br>Phases will be<br>included | EOS |
| 49 | ITT-E | Same shell as ARIA Week<br>48 Listing 49 | Listing of CD4+<br>Cell Count Data | Data in both<br>Phases will be<br>included | EOS |
| 50 | ITT-E | HIV4 | Listing of HIV-1<br>Associated<br>Conditions | Data in both<br>Phases will be<br>included | EOS |
| 51 | Safety | AE8 | Listing of Non-<br>Serious AEs of<br>Subjects at<br>Mexico sites | Mexican Safety Report requirement For EoS events in both phases will be included. | EOS |

| Non- | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 52 | Safety | AE8 | Listing of SAEs<br>of Subjects at<br>Mexico sites | Mexican Safety Report requirement For EoS events in both phases | EOS |
| 53 | Safety | AE8 | Listing of SAEs of Subjects at non-Mexico sites | will be included. Mexican Safety Report requirement For EoS events in both phases will be included. Include the country in one column | EOS |
| 65 | Safety-<br>Continuation<br>Phase | LIVER5 | Listing of Liver Event Results and Time of Event Relative to Treatment- Continuation Phase | | EOS |
| 69 | Safety | MH2 | Listing of Past<br>and Current Liver<br>Disease Medical<br>Conditions | | EOS |
| 70 | Safety-<br>Continuation<br>Phase | LB5 | Listing of Laboratory Data from Liver Event Follow-Up- Continuation Phase | | EOS |
| 71 | Safety-<br>Continuation<br>Phase | PREG1a | Listing of Subjects Who Became Pregnant During the Study- Continuation Phase | | EOS |

| Non- | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 82 | Safety-<br>Continuation<br>Phase | ECSSRS4 | Listing of C-<br>SSRS Suicidal<br>Ideation and<br>Behaviour Data-<br>Continuation<br>Phase | Add another column to show positive or negative. | EOS |
| 83 | Safety-<br>Continuation<br>Phase | PAN12 | Listing of COVID-19 Assessments and Symptom Assessments- Continuation Phase | New Output | EOS |
| 86 | Safety-<br>Continuation<br>Phase | Same as Listing 13 | Listing of Start<br>and Stop dates<br>in the<br>Continuation<br>Phase | New Output | EOS |
| 76 | ITT=E | Same shell as ARIA Week<br>48 Listing 76 | Listing of All<br>Genotypic Data | Both Randomized and Continuation Phase will be included in separate pages | EOS |
| 78 | ITT-E | Same shell as ARIA Week<br>48 Listing 78 | Listing of All<br>Phenotypic Data | Both Randomized and Continuation Phase will be included in separate pages | EOS |
| 84 | Genotypic<br>and/or<br>Phenotypic | /arenv/arprod/GSK1349572/<br>ING111762/ final_01/Listing<br>37 | Listing of Genotypic and Phenotypic Data for Subjects Meeting Confirmed Virologic Withdrawal Criteria | New Output; Both Randomized and Continuation Phase will be included in separate pages | EOS |

| Non- | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable |
| 85 | ITT-E | /arenv/arprod/GSK1349572/<br>ING111762/ final_01/Listing<br>38. | Listing of Genotypic and Phenotypic Data for Subjects with On-Treatment Virology Results at Non-CVW Timepoints | New Output; Both Randomized and Continuation Phase will be included in separate pages | EOS |

### 12.14. Appendix 14: List of Data Displays

### 12.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.n | 6.1 to 6.n |
| Virology | 7.1 to 7.n | NA |
| Section | List | ings |
| ICH Listings 1 to x | | |
| Other Listings | y to z | |

### 12.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 12.14.3. Deliverable

| Delivery | Description |
|----------|--------------------------------------------------|
| WK48 | Week 48 Statistical Analysis Complete |
| EOS | Final End of Study Statistical Analysis Complete |

# 12.14.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | <u>.</u> |
| 1.1. | All Subjects<br>Screened | SA1 | Summary of Study Populations | CS CORE; | WK48 |
| 1.2. | All Subjects<br>Screened | ES6 | Summary of Reasons for Screen Failure | CS CORE | WK48 |
| 1.3. | ITT(E) | EudraCT age | Summary of Age Categories | CS CORE | WK48 |
| 1.4. | ITT(E) | ES1 | Summary of Subject Accountability: Randomized Phase Conclusion Record | FDAAA, EudraCT | WK48 |
| 1.5. | ITT(E) | ES1 | Summary of Subject Accountability: Continuation Phase Conclusion Record | FDAAA, EudraCT | WK48 |
| 1.6. | ITT(E) | HIV_ES1 | Summary of Subject Accountability: Withdrawals by Visit | | WK48 |
| 1.7. | ITT(E) -<br>Continuation<br>Phase | DV1a | Summary of Important Protocol Deviations | CS CORE | WK48, EOS |
| 1.8. | ITT(E) | SA2 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | CS CORE | WK48 |
| Demog | raphy | | | | |
| 1.9. | ITT(E) | DM1 | Summary of Demographic Characteristics | CS CORE | WK48 |
| 1.10. | ITT(E) | DM5 | Summary of Race and Racial Combinations | CS CORE | WK48 |
| 1.11. | ITT(E) | DM6 | Summary of Race and Racial Combinations Details | CS CORE | WK48 |
| 1.12. | ITT(E) | | Summary of Hepatitis Status at Entry | | WK48 |
| 1.13. | ITT(E) | CDC1 | Summary of CDC Classification of HIV Infection at Baseline | | WK48 |

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.14. | ITT(E) | RF1 | Summary of HIV Risk Factors | | WK48 |
| 1.15. | ITT(E) | | Summary of Baseline Cardiovascular Risk Assessments | | WK48 |
| 1.16. | ITT(E) | | Distribution of Quantitative Plasma HIV-1 RNA Results at Screening and Baseline | | WK48 |
| 1.17. | ITT(E) | | Distribution of CD4+ Cell Count (cells/mm^3) Results at Screening and Baseline | | WK48 |
| Medica | l Conditions, C | oncomitant Medic | cations & ART | | |
| 1.18. | ITT(E) | MH1 | Summary of Current Medical Conditions | CS CORE | WK48 |
| 1.19. | ITT(E) | MH1 | Summary of Past Medical Conditions | CS CORE | WK48 |
| 1.20. | ITT(E) | MH4 | Summary of Current Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions | | WK48 |
| 1.21. | ITT(E) | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions | | WK48 |
| 1.22. | ITT(E) | CM1 | Summary of Concomitant Medication by Ingredient ATC Level 1 | | WK48 |
| 1.23. | ITT(E) | CM8 | Summary of Concomitant Medication Ingredient Combinations | | WK48 |
| 1.24. | ITT(E) | CM1b | Summary of Concomitant Medication by Combination Term ATC Level 1 | | WK48 |
| 1.25. | ITT(E) | | Summary of Lipid Modifying Agent Use at Baseline | | WK48 |
| 1.26. | ITT(E) | | Summary of Lipid Modifying Agent Use Starting Post-<br>Baseline | | WK48 |

| 3 | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| | No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1 | 1.27. | All Subjects<br>Screened | | Summary of Subjects by Country and Investigator | | WK48 |

# 12.14.5. Efficacy Tables

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Primary | Efficacy Anal | yses | | | |
| 2.1. | ITT(E) | | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 – Snapshot Analysis | | WK48 |
| 2.2. | Per-<br>Protocol | | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 – Snapshot Analysis | | WK48 |
| 2.3. | ITT | | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 – Snapshot Analysis | | WK48 |
| 2.4. | ITT(E) | | Summary of Study Outcomes (<50 c/mL) at Week 48 – Snapshot Analysis | | WK48 |
| 2.5. | ITT(E) | | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 - Snapshot Analysis | | WK48 |
| Second | ary Efficacy A | nalyses | | | |
| 2.6. | ITT(E) | | Summary of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 by Subgroup - Snapshot Analysis | | WK48 |
| 2.7. | ITT(E) | | Summary of Change from Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit | | WK48, EOS |
| 2.8. | ITT(E) | | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit – Snapshot Analysis | | WK48 |
| 2.9. | ITT(E) | | Proportion of Subjects with Plasma HIV-1 RNA <400 c/mL by Visit – Snapshot Analysis | | WK48 |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.10. | ITT(E) | | Summary of Study Outcomes (<400 c/mL) at Week 48 – Snapshot Analysis | | WK48 |
| 2.11. | ITT(E) | | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal at Week 48 - Treatment Related Discontinuation = Failure | | WK48 |
| 2.12. | ITT(E) | | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal at Week 48 - Efficacy Related Discontinuation = Failure | | WK48 |
| 2.13. | ITT(E) | Same shell as<br>ARIA Week 48 | Proportion of Subjects Meeting Confirmed Virologic Withdrawal Criteria by Visit- Observed Case | | WK48, EOS |
| 2.14. | ITT(E) | | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Withdrawal | | WK48 |
| 2.15. | ITT(E) | Same shell as<br>ARIA Week 48 | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit | | WK48, EOS |
| 2.16. | ITT(E) | HIV1 | Summary of Post-Baseline HIV-1 Associated Conditions Including Recurrences | | WK48, EOS |
| 2.17. | ITT(E) | HIV1 | Summary of Post-Baseline HIV-1 Associated Conditions Excluding Recurrences | | WK48, EOS |
| 2.18. | ITT(E) | HIV2 | Summary of Post-Baseline HIV-1 Disease Progressions | | WK48, EOS |
| 2.19. | ITT(E) | gsk2619619/<br>mid200336/<br>final_01/table<br>2.1 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit – Observed Case | | EOS |

## 12.14.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Insert E | ndpoint Categ | ory | | | |
| 2.1. | ITT(E) | | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit – Snapshot Analysis | Line plot | WK48 |
| 2.2. | ITT(E) | Same shell as<br>Gemini Figure<br>2.3 | Individual Plasma HIV-1 RNA (log10 c/mL) and CD4+ Profiles by Visit for Subjects with at least One Suspected Virologic Withdrawal Visit | | WK48, EOS |
| 2.3. | ITT(E) | | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week 48 by Subgroup – Snapshot Analysis | | WK48 |

## 12.14.7. Safety Figures

| Safety | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Insert E | Insert Endpoint Category | | | | |
| 3.1. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk | CS CORE | WK48 |
| 3.2. | Safety | LIVER9 | Scatter Plot of Maximum vs. Baseline for ALT | CS CORE | WK48 |
| 3.3. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | CS CORE | WK48, EOS |
| 3.4. | Safety | | Line Plot of mean change from Baseline in Creatinine | | WK48 |
| 3.5. | Safety | | Bar Chart of Triglycerides (mmol/L) NCEP Categories at Week 48 vs. Baseline | | WK48 |
| 3.6. | Safety | | Bar Chart of Total Cholesterol (mmol/L) NCEP Categories at Week 48 vs. Baseline | | WK48 |
| 3.7. | Safety | | Bar Chart of HDL Cholesterol (mmol/L) NCEP Categories at Week 48 vs. Baseline | | WK48 |
| 3.8. | Safety | | Bar Chart of LDL Cholesterol (mmol/L) NCEP Categories at Week 48 vs. Baseline | | WK48 |
| 3.9. | Safety | | Bar Chart of Total Cholesterol/ HDL Ratio at Week 48 vs. Baseline | | WK48 |

#### 12.14.8. Health Outcomes Tables

| Health | Health Outcomes : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| SF-12 | | | | | |
| 6.1. | ITTE | | Summary of SF-12 Individual Item Scores - LOCF | | WK48 |
| 6.2. | ITTE | | Summary of SF-12 Total score, MCS and PCS by Visit - LOCF | Results to go into summary stats come from a computer analysis progam | WK48 |
| 6.3. | ITTE | | Summary of SF-12 Total score, MCS and PCS by Visit - Observed | Results to go into summary stats come from a computer analysis progam | WK48 |
| 6.4. | ITTE | | Summary of Change from Baseline at Week 48 in SF-12 Total score, MCS and PCS - LOCF | Results to go into summary stats come from a computer analysis progam | WK48 |
| 6.5. | ITTE | | Summary of Change from Baseline at Week 48 in SF-12 Total score, MCS and PCS - Observed | Results to go into summary stats come from a computer analysis progam | WK48 |
| HIVTSO | Ìs | | | | |
| 6.6. | ITTE | | Summary of HIVTSQs Individual Item Scores by Visit - LOCF | | WK48 |
| 6.7. | ITTE | | Summary of HIVTSQs Total Score by Visit - LOCF | | WK48 |
| 6.8. | ITTE | | Summary of HIVTSQs Total Score by Visit - Observed | | WK48 |
| 6.9. | ITTE | | Summary of HIVTSQs Lifestyle/ease Sub-score by visit - LOCF | | WK48 |
| 6.10. | ITTE | | Summary of HIVTSQs Lifestyle/ease Sub-score by visit - Observed | | WK48 |
| 6.11. | ITTE | | Summary of HIVTSQs General Satisfaction/Clinical Sub-score by visit - LOCF | | WK48 |
| 6.12. | ITTE | | Summary of HIVTSQs General Satisfaction/Clinical Sub-score by visit - Observed | | WK48 |

## 12.14.9. Virology Tables

| Virolog | Virology : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Genoty | ре | | | | |
| 7.1. | Genotypic | | Summary of INI Mutations at time of CVW | | WK48 |
| 7.2. | Genotypic | | Summary of Treatment Emergent INI Mutations at time of CVW | | WK48 |
| 7.3. | Genotypic | | Summary of Major Mutations of NRTI, NNRTI and PI Classes at time of CVW | | WK48 |
| 7.4. | Genotypic | | Summary of Treatment Emergent Major Mutations of NRTI, NNRTI and PI Classes at time of CVW | | WK48 |
| Phenot | уре | | | | |
| 7.5. | Phenotypic | | Summary of Phenotype at time of CVW by phenotypic cut-<br>off | For EoS both phases will be included | WK48, EOS |
| 7.6. | Phenotypic | | Summary of Phenotype at time of CVW by Number of Drugs to Which Subject are Resistant | | WK48 |
| 7.7. | Phenotypic | | Summary of Fold Change at Baseline and Time of CVW | For EoS both phases will be included. | WK48, EOS |
| 7.8. | Phenotypic | | Summary of Change from Baseline in Fold Change at Time of CVW | | WK48 |

## 12.14.10. Safety Tables

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exposu | re | | | | • |
| 3.1. | Safety | | Summary of Extent of Exposure to Investigational Product - Randomised Phase | CS Core | WK48 |
| 3.2. | Safety | | Summary of Extent of Exposure to Investigational Product - Randomisation and Continuation Phase | CS Core | WK48, EOS |
| Adverse | Events | | | | |
| 3.3. | Safety | AE5 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity-Randomised Phase | CS Core | WK48, EOS |
| 3.4. | Safety | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency-Randomised Phase | CS Core | WK48, EOS |
| 3.5. | Safety | AE3 | Summary of Common (>=3%) Grade 2-4 Adverse Events by Overall Frequency-Randomised Phase | CS Core | WK48, EOS |
| 3.6. | Safety | AE5 | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Toxicity-Randomised Phase | CS Core | WK48, EOS |
| 3.7. | Safety | AE3 | Summary of Common (>=3%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency-Randomised Phase | CS Core | WK48, EOS |
| 3.8. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class – Randomised Phase | CS Core | WK48 |
| 3.9. | Safety | AE1 | Summary of Serious Adverse Events by System Organ<br>Class – Randomised and Continuation Phase | CS Core New output. FDAAA, EudraCT | WK48, EOS |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.10. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class-Randomised Phase | CS Core Plain Language Summary (PLS) requirements | WK48 |
| 3.11. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product – Randomised Phase | CS Core | WK48 |
| 3.12. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product – Randomised and Continuation Phase | CS Core | WK48, EOS |
| 3.13. | Safety | AE3 | Summary of Common (>=3%) Non-Serious Adverse Events-Randomised and Continuation Phase | CS Core<br>FDAAA | WK48, EOS |
| 3.14. | Safety | EudraCT Non-<br>serious AE | Summary of Subjects and Number of Occurrences of Common (>=3%) Non-Serious Adverse Events by System Organ Class-Randomised and Continuation Phase | CS Core<br>EudraCT | WK48, EOS |
| 3.15. | Safety | EudraCT SAE | Summary of Subjects and Number of occurrences of SAEs, Drug-related AEs, Fatal SAEs, and Drug-related SAEs-Randomised and Continuation Phase | CS Core<br>EudraCT | WK48, EOS |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | tory | | | | |
| 3.16. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit | CS Core | WK48 |
| 3.17. | Safety | LB1 | Summary of Lipids Percentage Changes from Baseline by Visit | | WK48 |
| 3.18. | Safety | LB1 | Summary of Hematology Changes From Baseline by Visit | CS Core | WK48 |
| 3.19. | Safety | LB1 | Summary of Urine Concentrations Changes from Baseline by Visit | CS Core | WK48 |
| 3.20. | Safety | | Summary of Maximum Post-Baseline in Urinalysis Dipstick Results | | WK48 |
| 3.21. | Safety | | Summary of Changes in Proteinuria Baseline Laboratory Result to Maximum Post-Baseline Laboratory Result - Randomised Phase | i.e., "shift table" | WK48 |
| 3.22. | Safety | | Summary of Changes in NCEP Lipid Baseline Category to Maximum Post-Baseline Category - Triglycerides Randomised Phase | | WK48 |
| 3.23. | Safety | | Summary of Changes in NCEP Lipid Baseline Category to Maximum Post-Baseline Category – Total Cholesterol Randomised Phase | | WK48 |
| 3.24. | Safety | | Summary of Changes in NCEP Lipid Baseline Category to Maximum Post-Baseline Category – HDL Cholesterol Randomised Phase | | WK48 |
| 3.25. | Safety | | Summary of Changes in NCEP Lipid Baseline Category to Maximum Post-Baseline Category – LDL Cholesterol Randomised Phase | | WK48 |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.26. | Safety | | Summary of TC/HDL ratio Changes from Baseline Randomised Phase | | WK48 |
| 3.27. | Safety | | Summary of Bone Markers Changes from Baseline Randomised Phase | | WK48 |
| 3.28. | Safety | | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities – Randomised Phase | CS Core | WK48 |
| 3.29. | Safety | | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities – Randomised and Continuation Phase | CS Core | WK48, EOS |
| 3.30. | Safety | | Summary of Maximum Post-Baseline Emergent Hematology Toxicities – Randomised Phase | CS Core | WK48 |
| 3.31. | Safety | | Summary of Maximum Post-Baseline Emergent Hematology Toxicities – Randomised and Continuation Phase | CS Core | WK48, EOS |
| 3.32. | Safety | | Statistical analysis of Change from Baseline in Triglycerides at Week 48 (Multiple imputed Dataset - MAR) | | WK48 |
| 3.33. | Safety | | Statistical analysis of Change from Baseline in Triglycerides at Week 48 - OC Dataset | | WK48 |
| 3.34. | Safety | | Statistical analysis of Change from Baseline in Triglycerides at Week 48 - Lipid LOCF Dataset | | WK48 |
| 3.35. | Safety | | Statistical analysis of Change from Baseline in<br>Triglycerides at Week 48 - Repeated Measures Mixed<br>Model Analysis | | WK48 |
| 3.36. | Safety | | Statistical analysis of Change from Baseline in TC/HDL<br>Ratio at Week 48 (Multiple imputed Dataset - MAR) | | WK48 |
| 3.37. | Safety | | Statistical analysis of Change from Baseline in TC/HDL<br>Ratio at Week 48 - Observed Case | | WK48 |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.38. | Safety | | Statistical analysis of Change from Baseline in TC/HDL<br>Ratio at Week 48 - Lipid LOCF | | WK48 |
| 3.39. | Safety | | Statistical analysis of Change from Baseline in TC/HDL<br>Ratio at Week 48 - Repeated Measures Mixed Model<br>Analysis | | WK48 |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Other | | | | | |
| 3.40. | Safety | ABC_HSR1 | Summary of the Incidence of Abacavir Hypersensitivity Reaction Classified as SAEs | Safety population, subset to those exposed to abacavir. Total column combines all treatment groups. | WK48 |
| 3.41. | Safety | OLIVER1 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria at Any Post-Baseline Visit | | WK48, EOS |
| 3.42. | Safety | | Subjects Meeting Hepatobiliary Abnormality Criteria - Post-<br>Baseline Emergent | | WK48, EOS |
| 3.43. | Safety | | Summary of Positive Suicidal indication Alerts based on eCSSRS by Visit | | WK48 |
| 3.44. | Safety | | Statistical Analysis of Bone Specific Alkaline Phosphatase (Ratio of Week 48 Result over Baseline) | | WK48 |
| 3.45. | Safety | | Statistical Analysis of Type I Collagen C-Telopeptides (Ratio of Week 48 Result over Baseline) | | WK48 |
| 3.46. | Safety | | Statistical Analysis of Osteocalcin (Ratio of Week 48 Result over Baseline) | | WK48 |
| 3.47. | Safety | | Statistical Analysis of Procollagen 1 N-Terminal Propeptide (Ratio of Week 48 Result over Baseline) | | WK48 |
| 3.48. | Safety | | Statistical Analysis of Vitamin D (Ratio of Week 48 Result over Baseline) | | WK48 |
| 3.49. | Safety | | Summary of All Adverse Events by System Organ Class - Randomised Phase | | WK48 |

# 12.14.11. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Study | Population | | | • | |
| 1. | Randomized | TA1 | Listing of Randomized and Actual Strata and Treatment Assignment | CS CORE | WK48 |
| 2. | All Subjects<br>Screened | ES7 | Listing of Reasons for Screen Failure | CS CORE | WK48 |
| 3. | Randomized | | Listing of Subjects Randomized But Not Treated | CS CORE (related to 'Listing for exclusion from any population) | WK48 |
| 4. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | CS CORE / | WK48, EOS |
| 5. | ITT-E | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | CS CORE | WK48 |
| 6. | ITT-E | | Listing of Important Protocol Deviations | CS CORE | WK48, EOS |
| 7. | ITT-E | | Listing of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | CS CORE (add listing for exclusion of other populations?) | WK48 |
| 8. | ITT-E | DM2 | Listing of Demographic Characteristics | CS CORE | WK48 |
| 9. | ITT-E | DM9 | Listing of Race | CS CORE | WK48 |
| Efficac | у | | | | |
| 10. | ITT-E | | Listing of Quantitative Plasma HIV-1 RNA Data | | WK48, EOS |
| 11. | ITT-E | | Listing of Study Outcome (<50 c/mL) at Week 48 – Snapshot Analysis | | WK48 |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 12. | ITT-E | | Listing of Study Outcome (<400 c/mL) at Week 48 – Snapshot Analysis | | WK48 |
| Safety | | | | | |
| 13. | Safety | HIV_IP5 | Listing of Investigational Product Exposure Data | CS CORE | WK48, EOS |
| 14. | Safety | | Listing of Investigational Product Exposure Data - Mexican Subjects | | WK48 |
| 15. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | CS CORE | WK48 |
| 16. | Safety | AE8 | Listing of All Adverse Events | CS CORE | WK48, EOS |
| 17. | Safety | AE8 | Listing of Fatal Adverse Events | CS CORE | WK48, EOS |
| 18. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | CS CORE | WK48, EOS |
| 19. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | CS CORE | WK48, EOS |
| 20. | Safety-<br>Continuation<br>Phase | AE2 | Listing of Relationship of Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | CS CORE For EoS only report events in the Continuation Phase; Add "-Continuation Phase to the title" | WK48, EOS |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 21. | Safety | SAE Reasons | Listing of Reasons for Considering as a Serious Adverse Event | CS CORE<br>FDA | WK48 |
| 22. | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data for Subjects with Laboratory Abnormalities of Potential Clinical Concern | CS CORE | WK48, EOS |
| 23. | Safety | LB5 | Listing of Hematology Laboratory Data for Subjects with Laboratory Abnormalities of Potential Clinical Concern | CS CORE | WK48 |
| 24. | Safety | UR2a | Listing of Urinalysis Data for Subjects with Abnormalities of Potential Clinical Concern | CS CORE | WK48 |
| 25. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data: Event and Description (Section 1- Section 2) | | WK48, EOS |
| 26. | Safety | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | | WK48, EOS |
| 27. | Safety | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | | WK48, EOS |
| 28. | Safety | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5- Section 8) | | WK48, EOS |

## 12.14.12. Non-ICH Listings

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | | | | |
| 29. | All Subjects<br>Screened | | Listing of Study Populations | | WK48, EOS |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 30. | All Subjects<br>Screened | | Listing of Subject Recruitment by Country and Site Number | | WK48 |
| 31. | All Subjects<br>Screened | | Listing of Rescreened Subjects | | WK48 |
| 32. | ITT-E | | Listing of Visit Dates | | WK48, EOS |
| 33. | ITT-E | | Listing of Hepatitis Test Results | | WK48 |
| 34. | ITT-E | CDC3 | Listing of CDC Classification of HIV Infection at Baseline | | WK48 |
| 35. | ITT-E | RF2 | Listing of HIV Risk Factors | | WK48 |
| 36. | ITT-E | MH2 | Listing of Current and Past Medical Conditions at Baseline | | WK48 |
| 37. | ITT-E | | Listing of Current and Past Medical Conditions at Baseline - Mexican subjects only | | WK48 |
| 38. | ITT-E | | Listing of Baseline Cardiovascular Risk Assessment Data | | WK48 |
| 39. | ITT-E | | Listing of History of Cardiac Therapeutic Procedures | | WK48 |
| 40. | ITT-E | | Listing of Investigational Product Accountability | | WK48, EOS |
| 41. | ITT-E | CM2 | Listing of Concomitant Medications | CS CORE | WK48, EOS |
| 42. | ITT-E | | Listing of Concomitant Medications - Mexican subjects only | | WK48 |
| 43. | ITT-E | CM6 | Listing of Relationship Between ATC Level 1, Ingredient and Verbatim Text | | WK48 |
| 44. | ITT-E | CM2 | Listing of Prior ART Medications | | WK48 |
| 45. | ITT-E | CM2 | Listing of Concomitant ART Medications | | WK48, EOS |
| 46. | ITT-E | | Listing of Concomitant ART Medications - Mexican subjects only | | WK48 |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 47. | ITT-E | CM6 | Listing of Relationship Between ATC Level 4, Ingredient and Verbatim Text | | WK48 |
| Efficac | у | | | | |
| 48. | ITT-E | Same shell as<br>ARIA Week 48 | Listing of Subjects with Confirmed Virologic Withdrawal | | WK48, EOS |
| 49. | ITT-E | Same shell as<br>ARIA Week 48 | Listing of CD4+ Cell Count Data | | WK48, EOS |
| 50. | ITT-E | HIV4 | Listing of HIV-1 Associated Conditions | | WK48, EOS |
| Safety | ı | 1 | | • | 1 |
| 51. | Safety | AE8 | Listing of Non-Serious AEs of Subjects at Mexico sites | Mexican Safety Report requirement For EoS events in both phases will be included. | WK48, EOS |
| 52. | Safety | AE8 | Listing of SAEs of Subjects at Mexico sites | Mexican Safety Report requirement | WK48, EOS |
| 53. | Safety | AE8 | Listing of SAEs of Subjects at non-Mexico sites | Mexican Safety Report requirement | WK48, EOS |
| 54. | Safety | AE8 | Listing of Pre-treatment Adverse Events | | WK48 |

| Non-ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 55. | Safety | | Listing of Cardiovascular Events | | WK48 |
| 56. | Safety | VS4 | Listing of Vital Signs | | WK48 |
| 57. | Safety | ABC_HSR<br>_EXPO2 | Listing of Abacavir Hypersensitivity Reaction Record - Exposure to Abacavir | | WK48 |
| 58. | Safety | ABC_HSR<br>_DRUG2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject History of Drug Allergies | | WK48 |
| 59. | Safety | ABC_HSR<br>COND2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject and Family Conditions | | WK48 |
| 60. | Safety | ABC_HSR<br>_RASH2 | Listing of Abacavir Hypersensitivity Reaction Record - Skin Rash Details | | WK48 |
| 61. | Safety | ABC_HSR<br>_SYMP4 | Listing of Abacavir Hypersensitivity Reaction Record - Symptoms | | WK48 |
| 62. | Safety | VS4 | Listing of Abacavir Hypersensitivity Reaction Record - Vital Signs | | WK48 |
| 63. | Safety | ABC_HSR<br>_SYMP6 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments (Excluding Other Symptoms) | | WK48 |
| 64. | Safety | ABC_HSR<br>_SYMP7 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments (Other Symptoms) | | WK48 |
| 65. | Safety | LIVER5 | Listing of Liver Event Results and Time of Event Relative to Treatment | | WK48, EOS |
| 66. | Safety | LIVER6 | Listing of Liver Event Information for RUCAM Score | | WK48 |
| 67. | Safety | LIVER7 | Listing of Liver Biopsy Details | | WK48 |
| 68. | Safety | LIVER8 | Listing of Liver Imaging Details | | WK48 |

| Non-ICI | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 69. | Safety | MH2 | Listing of Past and Current Liver Disease Medical Conditions | | WK48, EOS |
| 70. | Safety | LB5 | Listing of Laboratory Data from Liver Event Follow-Up | | WK48, EOS |
| 71. | Safety | PREG1a | Listing of Subjects Who Became Pregnant During the Study | | WK48, EOS |
| 72. | Safety | ECSSRS4 | Columbia Suicidality | | WK48, EOS |
| 81. | Safety | | Listing of Post Baseline Maximum ALT and Maximum Bilirubin - Randomised Phase | | WK48 |
| 82. | Safety | | Listing of Positive Suicidal Alerts Based on eCSSRS | | WK48 |
| Health ( | Outcomes | | | • | |
| 75. | ITT-E | | Listing of HIVTSQs | | WK48 |
| Pharma | cokinetic Anal | ysis | | | - 1 |
| 80. | Safety | | Listing of Pharmacokinetic Concentration Data | | WK48 |
| Virology | у | | | | |
| 76. | Genotypic | ARIA Week 48<br>Listing 76 | Listing of All Genotypic Data | Both Randomized and<br>Continuation Phase will be<br>included in separate pages | WK48, EOS |
| 77. | Genotypic | | Listing of Treatment Emergent Genotypic Mutations | | WK48 |
| 78. | Phenotypic | ARIA Week 48<br>Listing 78 | Listing of All Phenotypic Data | Both Randomized and<br>Continuation Phase will be<br>included in separate pages | WK48, EOS |

| Non-ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 79. | Phenotypic | | Listing of Replication Capacity | | WK48 |

# 12.15. Appendix 15: Example Mock Shells for Data Displays

Data display specifications will be uploaded as separate document.